CLINICAL TRIAL: NCT03639311
Title: A Phase IIb, Multicenter, Open-label, Rollover Study Evaluating the Efficacy, Safety and Tolerability of Long-acting Cabotegravir Plus Long-acting Rilpivirine Administered Every Two Months in HIV-1 Infected Adults Who Are Virologically Suppressed and Participated in Study LAI116482
Brief Title: Phase 2b, Open-label, Multicenter, Rollover Study to Assess Antiviral Activity and Safety of Long-acting (LA) Cabotegravir (CAB) Plus LA Rilpivirine (RPV), Administered Every 2 Months (Q2M), in Human Immunodeficiency Virus (HIV)-Positive Participants From the LATTE Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209035
Record Dates: First submitted 2018-08-10; First posted 2018-08-21 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: HIV; Antiretroviral therapy; Maintenance; Long acting; LATTE
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This is an Intervention Model, with parallel assignment, where the primary purpose of the study is, treatment, with 2 arms and no masking.
Masking Description: This is an open-label study, thus no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CAB LA + RPV LA Q2M (Experimental): Eligible participants from LAI116482 (NCT01641809 [LATTE]) study who were administered oral CAB 30 milligrams (mg) plus RPV 25 mg and who successfully completed Week 300 received their first dose CAB LA (600 mg) plus RPV LA (900 mg) injections within 2 hours of the final oral dose of LATTE given on the same day. The second loading injections were administered 1 month after initial loading dose, with subsequent injections (CAB LA 600 mg + RPV LA 900 mg) occurring Q2M thereafter. Participants continued to receive the treatment until the study intervention was locally approved and commercially available. Participants who received at least one dose of CAB LA and/or RPV LA and discontinued the CAB LA + RPV LA regimen for any reason entered a 52-week long-term follow-up (LTFU) Phase.
  Interventions: Drug: CAB LA; Drug: RPV LA
- DTG + RPV (Experimental): Eligible participants from LAI116482 (NCT01641809 [LATTE]) study who were administered oral CAB 30 mg plus RPV 25 mg and who successfully completed Week 300 received their first dose of the Dolutegravir (DTG) 50 mg plus RPV 25 mg, once daily as oral regimen on Day 1 until Month 12 in the current study. These participants were not eligible for the LTFU phase.
  Interventions: Drug: RPV; Drug: DTG
- LTFU: CAB LA+RPV LA Q2M Group (Experimental): This group included the participants who received at least one dose of CAB LA and/or RPV LA and discontinued the CAB LA + RPV LA regimen for any reason before end of Maintenance Period. The participants entered a 52-week LTFU period.
  Interventions: Drug: CAB LA; Drug: RPV LA

INTERVENTIONS:
Drug: CAB LA — Administered CAB LA (600 mg) Q2M, as intramuscular injection.
  Arms: CAB LA + RPV LA Q2M; LTFU: CAB LA+RPV LA Q2M Group
Drug: RPV LA — Administered RPV LA (900 mg), Q2M, as intramuscular injection.
  Arms: CAB LA + RPV LA Q2M; LTFU: CAB LA+RPV LA Q2M Group
Drug: RPV — Oral dose of RPV 25 mg, administered once daily from Day 1 up to Month 12
  Arms: DTG + RPV
Drug: DTG — Oral dose of DTG 50 mg administered once daily from Day 1 up to Month 12.
  Arms: DTG + RPV

SUMMARY:
This study (POLAR), is designed to assess the antiviral activity and safety of CAB LA plus RPV LA, administered Q2M, in approximately 100 adult HIV-1 infected, antiretroviral therapy (ART) experienced participants. Participants will rollover from the NCT01641809 (LATTE) study, who have completed minimum duration of Week 312 and with demonstrated HIV-1 ribonucleic acid (RNA) suppression (less than [<]50 copies (c) per milliliter [mL]), while receiving a two-drug regimen consisting of once-daily oral CAB at 30 milligram (mg) plus RPV at 25 mg. The participants will be offered the option to switch to the LA, intramuscular injections of CAB LA plus RPV LA, Q2M or the oral fixed dose combination (FDC) of dolutegravir (DTG) plus RPV, for the continued maintenance of HIV-1 RNA suppression, known as the Maintenance Phase (From Day 1 to Commercial Approval). Duration of study will vary from country to country, until regimen receives regulatory approval and becomes commercially available. The study plans to enroll approximately 100 participants. Any participant who receives at least one dose of CAB LA and/or RPV LA and discontinues the CAB LA plus RPV LA regimen for any reason will enter a 52-week Long-Term Follow-Up (LTFU) phase. Those participants must remain on suppressive highly active antiretroviral therapy (HAART) for at least 52 weeks after the last dose of CAB LA and or RPV LA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older (or >=19 where required by local regulatory agencies), at the time of signing the informed consent.
* A female participant is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test at Day 1), not lactating, and at least with one of following conditions:

  (a) Non-reproductive potential defined as: (i) Pre-menopausal females with one of the conditions as documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.

(ii) Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.

(b) Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication, throughout the study, for at least 30 days after discontinuation of all oral study medications, and for at least 52 weeks after discontinuation of CAB LA and RPV LA.

* The investigator is responsible for ensuring that participants understand how to properly use the methods of contraception.
* Capable of giving signed informed consent.
* Must have been on oral CAB 30 mg plus RPV 25 mg regimen through at minimum Week 300 of the LATTE study as per LATTE protocol dosing requirements and until Day 1 of the POLAR study. Any disruptions in dosing during LATTE must be discussed with the Medical Monitor for a final determination of eligibility.
* Plasma HIV-1 RNA <50 c/mL at Week 300. If participant has plasma HIV-1 RNA >= 50 c/mL at Week 300 in LATTE, a single repeat to determine eligibility may be allowed ONLY after consultation with the medical monitor.

Exclusion Criteria:

* During the last 6 months of participation in LATTE, consecutive (2 or more sequential) plasma HIV-1 RNA measurements >=50 c/mL.
* During the last 6 months of participation in LATTE, any HIV-1 RNA measurement >=200 c/mL.
* Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease [CDC, 2014], except cutaneous Kaposi's sarcoma not requiring systemic therapy.
* Participants with moderate to severe hepatic impairment determined by Child-Pugh classification.
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrolment if the Investigator believes the risk of seizure recurrence is low.
* Participants who, in the investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* Participants has a tattoo or other dermatological condition overlying the gluteus region which may interfere with interpretation of injection site reactions.
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV DNA as follows; Participants positive for HBsAg are excluded; participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded.
* Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Investigators must carefully assess if therapy specific for HCV infection is required; participants who are anticipated to require HCV treatment within 12 months must be excluded. (HCV treatment on study may be permitted, following consultation with the medical monitor).
* Participants with HCV co-infection will be allowed entry into this study if: Liver enzymes meet entry criteria; HCV Disease has undergone appropriate work-up, and is not advanced.
* Additional information (where available) on participants, with HCV co-infection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.
* In the event that recent biopsy or imaging data is not available or inconclusive, the fibrosis- 4 (Fib-4) score will be used to verify eligibility where Fib-4 score >3.25 is exclusionary; Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation where the Fibrosis 4 Score Formula: age multiplied by aspartate amino transferase (AST) divided by platelets multiplied by square of alanine aminotransferase (ALT).
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Ongoing or clinically relevant pancreatitis.
* Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the Study medical monitor for inclusion of the participant prior to randomization.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic (PK) sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
* Current or anticipated need for chronic anti-coagulation with the exception of the use of low dose acetylsalicylic acid (less than or equal to [<=]325 mg) or hereditary coagulation and platelet disorders such as hemophilia or Von Willebrand Disease.
* Corrected QT interval (QTc (Bazett)) >450 millisecond (msec) or QTc (Bazett) >480 msec for participants with bundle branch block.
* Any verified Grade 4 laboratory abnormality over the last 6 months in LATTE. A single repeat test is allowed to verify a result.
* Any acute laboratory abnormality over the last 6 months in LATTE, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
* ALT>=5 times upper limit of normal (ULN) or ALT >= 3 times ULN and bilirubin >= 1.5 times ULN (with >35 percent [%] direct bilirubin) over the last 6 months in LATTE.
* Exposure to an experimental drug (with the exception of those in the LATTE study including CAB and RPV) or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to Day 1 of this study.
* Treatment with any of the following agents within 28 days of Day 1: radiation therapy, cytotoxic chemotherapeutic agents, tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid [INH]); anti-coagulation agents.
* Immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons.
* Use of medications which are associated with Torsade de Pointes must be discussed with the Medical Monitor to determine eligibility.
* Participants receiving any prohibited medication and who are unwilling or unable to switch to an alternate medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (26):
- United States (23):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Macon, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Annandale, Virginia
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available, within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided, after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided, for an initial period of 12 months but an extension can be granted, when justified for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Okesanya OJ, Ayeni RA, Amadin P, Ngwoke I, Amisu BO, Ukoaka BM, Ahmed MM, Oso TA, Musa SS, Lucero-Prisno DE. Advances in HIV Treatment and Vaccine Development: Emerging Therapies and Breakthrough Strategies for Long-Term Control. AIDS Res Treat. 2025 Jul 4;2025:6829446. doi: 10.1155/arat/6829446. eCollection 2025. PMID 40655875
- [Derived] Mills A, Richmond GJ, Newman C, Osiyemi O, Cade J, Brinson C, De Vente J, Margolis DA, Sutton KC, Wilches V, Hatch S, Roberts J, McCoig C, Garris C, Vandermeulen K, Spreen WR. Long-acting cabotegravir and rilpivirine for HIV-1 suppression: switch to 2-monthly dosing after 5 years of daily oral therapy. AIDS. 2022 Feb 1;36(2):195-203. doi: 10.1097/QAD.0000000000003085. PMID 34652287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, open-label, rollover study evaluating the efficacy, safety and tolerability of long acting (LA) cabotegravir (CAB) plus LA rilpivirine (RPV) administered every 2 months (Q2M) in human immunodeficiency virus-1 (HIV-1) adult participants who were virologically suppressed and participated in study LAI116482 (NCT01641809).
Pre-assignment Details: This study was conducted in 2 phases (Maintenance Phase and Long-term Follow-up [LTFU] Phase). Maintenance Phase was defined from Baseline (Day 1) up to Month 52. LTFU Phase was defined as approximately 12 months for participants who discontinued from the CAB LA+RPV LA treatment before Month 52 and complied with protocol-defined criteria for withdrawal. Participants in both the phases were mutually inclusive.
Period: Maintenance Phase
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV | LTFU: CAB LA+RPV LA Q2M Group
Started | 90 | 7 | 0
Completed | 76 | 7 | 0
Not Completed | 14 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — DECISION BY SUBJECT OR PROXY | 7 | 0 | 0
Not completed — STUDY SITE TERMINATED BY SPONSOR | 3 | 0 | 0
Not completed — SUBJECT REACHED PROTOCOL-DEFINED STOPPING CRITERIA | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Period: Long-term Follow-up Phase (LTFU Phase)
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV | LTFU: CAB LA+RPV LA Q2M Group
Started (70 participants from CAB LA + RPV LA Q2M arm who completed the Maintenance Phase did not enter LTFU Phase as they completed the study and transitioned off CAB LA + RPV LA Q2M regimen to other options. DTG + RPV arm was not considered for LTFU Phase.) | 0 | 0 | 6
Completed (70 participants from CAB LA + RPV LA Q2M arm who completed the Maintenance Phase did not enter LTFU Phase as they completed the study and transitioned off CAB LA + RPV LA Q2M regimen to other options. DTG + RPV arm was not considered for LTFU Phase.) | 0 | 0 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV | Total
Number analyzed (Participants) | 90 | 7 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Overall Study | 41.2 (9.49) | 49.1 (11.42) | 41.7 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 88 | 7 | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian-Japanese/East Asian/South East Asian Heritage | 1 | 0 | 1
  Black or African American | 21 | 3 | 24
  White | 63 | 4 | 67
  Multiple | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-ribonucleic Acid (RNA) >=50 Copies Per Milliliter (c/mL) as Per Food and Drug Administration (FDA) Snapshot Algorithm at Month 12 [Maintenance Phase]
Description: Percentage of participants with HIV-1 RNA >=50 c/mL as per FDA snapshot algorithm at Month 12 was assessed to demonstrate the antiviral activity of CAB LA+RPV LA Q2M and DTG + RPV regimen in HIV-1 infected antiretroviral therapy (ART) experienced participants. The HIV-1 RNA >=50 c/mL per Snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the 12 months analysis visit window.
Time Frame: At Month 12 [Maintenance Phase]
Population: Intent-to-treat-Exposed (ITT-E) population comprised of all participants who received at least one dose of investigational product (IP) during on or after Day 1 visit. Participants were analyzed according to the selected treatment regardless of what treatment was actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Percentage of participants | 0 [0.0 to 4.0] | 0 [0.0 to 41.0]

2. Secondary Outcome: Percentage of Participants With HIV-RNA <50 c/mL as Per FDA Snapshot Algorithm at Month 12 [Maintenance Phase]
Description: Percentage of participants with HIV-1 RNA <50 c/mL as per FDA snapshot algorithm at Month 12 was assessed to demonstrate the antiviral activity of CAB LA+RPV LA Q2M and oral DTG + RPV regimen. The HIV-1 RNA <50 c/mL per Snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the 12 months analysis visit window.
Time Frame: At Month 12 [Maintenance Phase]
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Percentage of participants | 98 [95 to 100] | 100 [59 to 100]

3. Secondary Outcome: Number of Participants With Protocol-defined Confirmed Virologic Failure up to End of Maintenance Phase
Description: Confirmed virologic failure was defined as rebound as indicated by two consecutive plasma HIV-1-RNA levels >=200 c/mL after prior suppression to <200 c/mL.
Time Frame: Up to End of Maintenance Phase (up to Month 52 for CAB LA+RPV LA Q2M group, up to Month 12 for DTG+RPV group)
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Participants | 1 | 0

4. Secondary Outcome: Percentage of Participants With HIV-RNA >=50 c/mL as Per FDA Snapshot Algorithm Over Time for CAB LA + RPV LA Q2M Arm up to Month 12 [Maintenance Phase]
Description: Percentage of participants with HIV-1 RNA >=50 c/mL as per FDA snapshot algorithm over time was assessed to demonstrate the antiviral activity of CAB LA+RPV LA Q2M regimen in HIV-1 infected ART experienced participants. The HIV-1 RNA >=50 c/mL per Snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the 12 months analysis visit window. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Baseline (Day 1) and at Months 2, 4, 6, 8, 10 and 12 [Maintenance Phase]
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAB LA + RPV LA Q2M
Number analyzed (Participants) | 90
Percentage of participants
  Baseline (Day 1) | 0 [0.0 to 4.0]
  Month 2 | 0 [0.0 to 4.0]
  Month 4 | 1 [0.0 to 3.3]
  Month 6 | 0 [0.0 to 4.0]
  Month 8 | 0 [0.0 to 4.0]
  Month 10 | 0 [0.0 to 4.0]
  Month 12 | 0 [0.0 to 4.0]

5. Secondary Outcome: Percentage of Participants With HIV-RNA >=50 c/mL as Per FDA Snapshot Algorithm Over Time for DTG + RPV up to Month 12 [Maintenance Phase]
Description: Percentage of participants with HIV-1 RNA >=50 c/mL as per FDA snapshot algorithm over time was assessed to demonstrate the antiviral activity of DTG + RPV regimen in HIV-1 infected ART experienced participants. The HIV-1 RNA >=50 c/mL per Snapshot algorithm was determined by the last on-treatment HIV-1 RNA measurement within the 12 months analysis visit window. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Baseline (Day 1) and at Months 3, 6, 9 and 12 [Maintenance Phase]
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Percentage of participants
  Baseline (Day 1) | 0.0 [0.0 to 41.0]
  Month 3 | 0.0 [0.0 to 41.0]
  Month 6 | 0.0 [0.0 to 41.0]
  Month 9 | 0.0 [0.0 to 41.0]
  Month 12 | 0.0 [0.0 to 41.0]

6. Secondary Outcome: Absolute Values for HIV-1 RNA of CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log10) values for plasma HIV-1 RNA have been presented. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Standard Deviation (SD)=0.0000 is defined as SD resulted below the detectable limit of the assay and approximate to 0.0000.
Time Frame: From Baseline (Day 1) up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase)
Population: ITT-E Population. Only those participants with data available for specific analysis and specified time points analyzed.
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Log 10 copies per milliliter
  Baseline (Day 1): number analyzed (Participants) | 89 | 0
  Baseline (Day 1) | 1.591 (0.0085) |
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | 1.590 (0.0000) |
  Month 4: number analyzed (Participants) | 89 | 0
  Month 4 | 1.594 (0.0305) |
  Month 6: number analyzed (Participants) | 89 | 0
  Month 6 | 1.590 (0.0042) |
  Month 8: number analyzed (Participants) | 89 | 0
  Month 8 | 1.590 (0.0000) |
  Month 10: number analyzed (Participants) | 88 | 0
  Month 10 | 1.594 (0.0384) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | 1.590 (0.0000) |
  Month 14: number analyzed (Participants) | 86 | 0
  Month 14 | 1.593 (0.0216) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | 1.598 (0.0555) |
  Month 18: number analyzed (Participants) | 85 | 0
  Month 18 | 1.592 (0.0217) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | 1.592 (0.0153) |
  Month 22: number analyzed (Participants) | 84 | 0
  Month 22 | 1.590 (0.0000) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | 1.602 (0.0882) |
  Month 26: number analyzed (Participants) | 85 | 0
  Month 26 | 1.611 (0.1246) |
  Month 28: number analyzed (Participants) | 86 | 0
  Month 28 | 1.594 (0.0334) |
  Month 30: number analyzed (Participants) | 83 | 0
  Month 30 | 1.590 (0.0000) |
  Month 32: number analyzed (Participants) | 84 | 0
  Month 32 | 1.590 (0.0000) |
  Month 34: number analyzed (Participants) | 84 | 0
  Month 34 | 1.590 (0.0000) |
  Month 36: number analyzed (Participants) | 82 | 0
  Month 36 | 1.590 (0.0000) |
  Month 38: number analyzed (Participants) | 80 | 0
  Month 38 | 1.590 (0.0000) |
  Month 40: number analyzed (Participants) | 78 | 0
  Month 40 | 1.590 (0.0000) |
  Month 42: number analyzed (Participants) | 78 | 0
  Month 42 | 1.590 (0.0000) |
  Month 44: number analyzed (Participants) | 75 | 0
  Month 44 | 1.591 (0.0104) |
  Month 46: number analyzed (Participants) | 69 | 0
  Month 46 | 1.590 (0.0000) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | 1.590 (0.0025) |
  Month 50: number analyzed (Participants) | 47 | 0
  Month 50 | 1.590 (0.0000) |
  Month 52: number analyzed (Participants) | 8 | 0
  Month 52 | 1.590 (0.0000) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | 1.852 (0.4338)
  LTFU Month 3: number analyzed (Participants) | 0 | 6
  LTFU Month 3 |  | 1.590 (0.0000)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | 1.590 (0.0000)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | 2.027 (1.0696)
  LTFU Month 12: number analyzed (Participants) | 0 | 6
  LTFU Month 12 |  | 1.616 (0.0581)

7. Secondary Outcome: Absolute Values for HIV-1 RNA of DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Logarithm to base 10 (log10) values for plasma HIV-1 RNA has been presented. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. SD=0.0000 is defined as SD resulted below the detectable limit of the assay and approximate to 0.0000.
Time Frame: At Baseline (Day 1) and at Months 3, 6, 9 and 12 [Maintenance Phase]
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Log 10 copies per milliliter
  Baseline (Day 1) | 1.590 (0.0000)
  Month 3 | 1.590 (0.0000)
  Month 6 | 1.590 (0.0000)
  Month 9 | 1.590 (0.0000)
  Month 12 | 1.590 (0.0000)

8. Secondary Outcome: Change From Baseline in HIV-1 RNA for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. Log 10 values for plasma HIV-1 RNA has been presented. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from baseline value is defined as post-dose value minus baseline value. SD=0.0000 is defined as SD resulted below the detectable limit of the assay and approximate to 0.0000.
Time Frame: Up to End of LTFU Phase (compared with Baseline [Day1]), (approximately up to 12 months after exiting the Maintenance Phase)
Population: ITT-E Population. Only those participants with data available for specific analysis and specified time points analyzed.
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Log 10 copies per milliliter
  Month 2: number analyzed (Participants) | 89 | 0
  Month 2 | -0.001 (0.0085) |
  Month 4: number analyzed (Participants) | 88 | 0
  Month 4 | 0.003 (0.0299) |
  Month 6: number analyzed (Participants) | 88 | 0
  Month 6 | -0.000 (0.0096) |
  Month 8: number analyzed (Participants) | 88 | 0
  Month 8 | -0.001 (0.0085) |
  Month 10: number analyzed (Participants) | 87 | 0
  Month 10 | 0.003 (0.0396) |
  Month 12: number analyzed (Participants) | 87 | 0
  Month 12 | -0.001 (0.0086) |
  Month 14: number analyzed (Participants) | 86 | 0
  Month 14 | 0.002 (0.0234) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | 0.007 (0.0529) |
  Month 18: number analyzed (Participants) | 85 | 0
  Month 18 | 0.001 (0.0235) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | 0.001 (0.0177) |
  Month 22: number analyzed (Participants) | 84 | 0
  Month 22 | -0.001 (0.0087) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | 0.011 (0.0888) |
  Month 26: number analyzed (Participants) | 85 | 0
  Month 26 | 0.020 (0.1251) |
  Month 28: number analyzed (Participants) | 86 | 0
  Month 28 | 0.003 (0.0346) |
  Month 30: number analyzed (Participants) | 83 | 0
  Month 30 | -0.001 (0.0088) |
  Month 32: number analyzed (Participants) | 84 | 0
  Month 32 | -0.001 (0.0087) |
  Month 34: number analyzed (Participants) | 84 | 0
  Month 34 | -0.001 (0.0087) |
  Month 36: number analyzed (Participants) | 82 | 0
  Month 36 | -0.001 (0.0088) |
  Month 38: number analyzed (Participants) | 80 | 0
  Month 38 | 0.000 (0.0000) |
  Month 40: number analyzed (Participants) | 78 | 0
  Month 40 | -0.001 (0.0091) |
  Month 42: number analyzed (Participants) | 78 | 0
  Month 42 | -0.001 (0.0091) |
  Month 44: number analyzed (Participants) | 75 | 0
  Month 44 | 0.000 (0.0140) |
  Month 46: number analyzed (Participants) | 69 | 0
  Month 46 | -0.001 (0.0096) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | -0.001 (0.0102) |
  Month 50: number analyzed (Participants) | 47 | 0
  Month 50 | 0.000 (0.0000) |
  Month 52: number analyzed (Participants) | 8 | 0
  Month 52 | 0.000 (0.0000) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | 0.262 (0.4338)
  LTFU Month 3: number analyzed (Participants) | 0 | 5
  LTFU Month 3 |  | 0.000 (0.0000)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | 0.000 (0.0000)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | 0.437 (1.0696)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | 0.026 (0.0581)

9. Secondary Outcome: Change From Baseline in HIV-1 RNA for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 8
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: Log 10 copies per milliliter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Log 10 copies per milliliter
  Month 3 | 0.000 (0.0000)
  Month 6 | 0.000 (0.0000)
  Month 9 | 0.000 (0.0000)
  Month 12 | 0.000 (0.0000)

10. Secondary Outcome: Absolute Values for Cluster of Differentiation 4 Plus (CD4+) for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity of CAB LA+RPV LA Q2M. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: From Baseline (Day 1) up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase)
Population: ITT-E Population. Only those participants with data available for specific analysis and specified time points analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Cells per cubic millimeter
  Baseline (Day 1): number analyzed (Participants) | 90 | 0
  Baseline (Day 1) | 873.0 (233.37) |
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | 868.1 (261.49) |
  Month 4: number analyzed (Participants) | 88 | 0
  Month 4 | 879.8 (280.88) |
  Month 6: number analyzed (Participants) | 5 | 0
  Month 6 | 1046.8 (435.74) |
  Month 8: number analyzed (Participants) | 88 | 0
  Month 8 | 857 (277.46) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | 859.2 (283.23) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | 917.5 (295.27) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | 912.8 (262.40) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | 910.3 (286.21) |
  Month 26: number analyzed (Participants) | 36 | 0
  Month 26 | 905.9 (274.22) |
  Month 28: number analyzed (Participants) | 84 | 0
  Month 28 | 867.3 (266.36) |
  Month 30: number analyzed (Participants) | 11 | 0
  Month 30 | 931.1 (220.94) |
  Month 32: number analyzed (Participants) | 82 | 0
  Month 32 | 853.7 (280.49) |
  Month 34: number analyzed (Participants) | 4 | 0
  Month 34 | 967.3 (300.72) |
  Month 36: number analyzed (Participants) | 80 | 0
  Month 36 | 865.4 (225.93) |
  Month 40: number analyzed (Participants) | 76 | 0
  Month 40 | 925.7 (271.70) |
  Month 42: number analyzed (Participants) | 4 | 0
  Month 42 | 1220.8 (536.73) |
  Month 44: number analyzed (Participants) | 76 | 0
  Month 44 | 905.7 (292.61) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | 1011.0 (292.74) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | 818.5 (291.82) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | 755.0 (182.43) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | 716.3 (143.21) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | 837.2 (224.49)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | 717.8 (188.88)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | 766.5 (184.84)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | 775.0 (293.45)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | 954.8 (259.47)

11. Secondary Outcome: Absolute Values for CD4+ for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity of DTG + RPV arm. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: At Baseline (Day 1) and at Months 3, 6, 9 and 12 [Maintenance Phase]
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Cells per cubic millimeter
  Baseline (Day 1) | 804.3 (167.73)
  Month 3 | 780.3 (145.22)
  Month 6 | 728.9 (147.06)
  Month 9 | 777.0 (251.37)
  Month 12 | 790.4 (141.80)

12. Secondary Outcome: Change From Baseline Values for CD4+ for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity of CAB LA+RPV LA Q2M. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from baseline value is defined as post-dose value minus baseline value.
Time Frame: as for outcome 8
Population: ITT-E Population. Only those participants with data available for specific analysis and specified time points analyzed.
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Cells per cubic millimeter
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | -4.9 (196.47) |
  Month 4: number analyzed (Participants) | 88 | 0
  Month 4 | 5.3 (221.68) |
  Month 6: number analyzed (Participants) | 5 | 0
  Month 6 | 100.2 (343.66) |
  Month 8: number analyzed (Participants) | 88 | 0
  Month 8 | -20.7 (218.39) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | -19.4 (189.19) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | 45.6 (227.11) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | 43.8 (193.72) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | 41.6 (224.99) |
  Month 26: number analyzed (Participants) | 36 | 0
  Month 26 | 4.2 (160.08) |
  Month 28: number analyzed (Participants) | 84 | 0
  Month 28 | -6.2 (196.62) |
  Month 30: number analyzed (Participants) | 11 | 0
  Month 30 | 18.1 (192.09) |
  Month 32: number analyzed (Participants) | 82 | 0
  Month 32 | -13.5 (215.60) |
  Month 34: number analyzed (Participants) | 4 | 0
  Month 34 | 15.8 (239.28) |
  Month 36: number analyzed (Participants) | 80 | 0
  Month 36 | 0.0 (195.92) |
  Month 40: number analyzed (Participants) | 76 | 0
  Month 40 | 67.1 (205.26) |
  Month 42: number analyzed (Participants) | 4 | 0
  Month 42 | 390.8 (406.79) |
  Month 44: number analyzed (Participants) | 76 | 0
  Month 44 | 31.6 (244.33) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | -98.5 (424.97) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | -44.2 (236.71) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -451.0 (485.08) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -23.0 (78.28) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -88.8 (156.64)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | -97.8 (188.52)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -111.8 (236.26)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -103.3 (87.22)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | 28.8 (209.33)

13. Secondary Outcome: Change From Baseline Values for CD4+ for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: Blood samples were collected and CD4+ cell count assessment by flow cytometry was carried out to evaluate the immunologic activity of DTG + RPV arm. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from baseline value is defined as post-dose value minus baseline value.
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: ITT-E Population
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Cells per cubic millimeter
  Month 3 | -24.0 (118.40)
  Month 6 | -75.4 (123.71)
  Month 9 | -27.3 (150.96)
  Month 12 | -13.9 (145.76)

14. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs >=5 Percent [%] Incidence) and Serious Adverse Events (SAEs) for CAB LA + RPV LA Q2M Arm
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement.
Time Frame: Up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase)
Population: Safety Population comprised of all participants who received at least one dose of study treatment on or after Day 1 visit. Participants were assessed according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M
Number analyzed (Participants) | 90
Participants
  Non-SAE (>=5%) | 86
  SAE | 10

15. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs >=5 Percent [%] Incidence) and Serious Adverse Events (SAEs) for DTG + RPV Arm
Description: as for outcome 14
Time Frame: Up to Month 12 [Maintenance Phase]
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Participants
  Non-SAE (>=5%) | 3
  SAE | 0

16. Secondary Outcome: Number of Participants With Severity of Adverse Events for CAB LA + RPV LA Q2M Arm
Description: Severity of adverse events were defined as per The Division of Acquired Immunodeficiency Syndrome (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS adverse events Grading Table). Severity grades for adverse events were Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Potentially life-threatening) and Grade 5 (all deaths related to an AE).
Time Frame: Up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M
Number analyzed (Participants) | 90
Participants
  Grade 1 | 22
  Grade 2 | 53
  Grade 3 | 10
  Grade 4 | 4
  Grade 5 | 0

17. Secondary Outcome: Number of Participants With Severity of Adverse Events for DTG + RPV Arm
Description: as for outcome 16
Time Frame: Up to Month 12 [Maintenance Phase]
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Participants
  Grade 1 | 0
  Grade 2 | 3
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

18. Secondary Outcome: Number of Participants With Maximum Post-Baseline Chemistry Toxicities for CAB LA + RPV LA Q2M Arm up to End of Maintenance Phase
Description: Clinical chemistry toxicities were graded as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table). Blood samples were collected for the analysis of following clinical chemistry parameters: alanine aminotransferase (ALT), albumin, aspartate aminotransferase (AST), bilirubin, carbon dioxide (CO2), cholesterol, creatinine kinase, creatinine, direct bilirubin, glomerular filtration rate (GFR) from creatinine adjusted using chronic kidney disease epidemiology collaboration (CKD-EPI), GFR from creatinine adjusted for bovine serum albumin (BSA), glucose, low density lipoprotein (LDL) cholesterol calculation, lipase, phosphate, sodium and triglycerides. Severity grades were: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening).
Time Frame: Up to End of Maintenance Phase (up to Month 52)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M
Number analyzed (Participants) | 90
Participants
  ALT, Grade 1 | 15
  ALT, Grade 2 | 3
  ALT, Grade 3 | 3
  ALT, Grade 4 | 0
  AST, Grade 1 | 12
  AST, Grade 2 | 6
  AST, Grade 3 | 0
  AST, Grade 4 | 0
  Bilirubin, Grade 1 | 4
  Bilirubin, Grade 2 | 1
  Bilirubin, Grade 3 | 0
  Bilirubin, Grade 4 | 0
  CO2, Grade 1 | 13
  CO2, Grade 2 | 0
  CO2, Grade 3 | 0
  CO2, Grade 4 | 0
  Cholesterol, Grade 1 | 8
  Cholesterol, Grade 2 | 5
  Cholesterol, Grade 3 | 0
  Cholesterol, Grade 4 | 0
  Creatine kinase, Grade 1 | 8
  Creatine kinase, Grade 2 | 7
  Creatine kinase, Grade 3 | 6
  Creatine kinase, Grade 4 | 2
  Creatinine, Grade 1 | 3
  Creatinine, Grade 2 | 0
  Creatinine, Grade 3 | 0
  Creatinine, Grade 4 | 0
  Direct bilirubin, Grade 1 | 0
  Direct bilirubin, Grade 2 | 0
  Direct bilirubin, Grade 3 | 1
  Direct bilirubin, Grade 4 | 0
  GFR from creatinine adjusted using CKD-EPI, Grade 1 | 0
  GFR from creatinine adjusted using CKD-EPI, Grade 2 | 23
  GFR from creatinine adjusted using CKD-EPI, Grade 3 | 3
  GFR from creatinine adjusted using CKD-EPI, Grade 4 | 0
  GFR from creatinine adjusted for BSA, Grade 1 | 0
  GFR from creatinine adjusted for BSA, Grade 2 | 23
  GFR from creatinine adjusted for BSA, Grade 3 | 3
  GFR from creatinine adjusted for BSA, Grade 4 | 0
  Glucose, Grade 1 | 21
  Glucose, Grade 2 | 20
  Glucose, Grade 3 | 0
  Glucose, Grade 4 | 0
  LDL cholesterol calculation, Grade 1 | 7
  LDL cholesterol calculation, Grade 2 | 4
  LDL cholesterol calculation, Grade 3 | 1
  LDL cholesterol calculation, Grade 4 | 0
  Lipase, Grade 1 | 10
  Lipase, Grade 2 | 15
  Lipase, Grade 3 | 3
  Lipase, Grade 4 | 4
  Phosphate, Grade 1 | 14
  Phosphate, Grade 2 | 2
  Phosphate, Grade 3 | 0
  Phosphate, Grade 4 | 0
  Sodium, Grade 1 | 9
  Sodium, Grade 2 | 1
  Sodium, Grade 3 | 0
  Sodium, Grade 4 | 0
  Triglycerides, Grade 1 | 11
  Triglycerides, Grade 2 | 8
  Triglycerides, Grade 3 | 2
  Triglycerides, Grade 4 | 1

19. Secondary Outcome: Number of Participants With Maximum Post-Baseline Chemistry Toxicities for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 18
Time Frame: Up to Month 12 [Maintenance Phase]
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Participants
  ALT, Grade 1 | 1
  ALT, Grade 2 | 0
  ALT, Grade 3 | 0
  ALT, Grade 4 | 0
  AST, Grade 1 | 0
  AST, Grade 2 | 0
  AST, Grade 3 | 0
  AST, Grade 4 | 0
  Bilirubin, Grade 1 | 0
  Bilirubin, Grade 2 | 0
  Bilirubin, Grade 3 | 0
  Bilirubin, Grade 4 | 0
  CO2, Grade 1 | 1
  CO2, Grade 2 | 0
  CO2, Grade 3 | 0
  CO2, Grade 4 | 0
  Cholesterol, Grade 1 | 0
  Cholesterol, Grade 2 | 0
  Cholesterol, Grade 3 | 0
  Cholesterol, Grade 4 | 0
  Creatine kinase, Grade 1 | 0
  Creatine kinase, Grade 2 | 0
  Creatine kinase, Grade 3 | 0
  Creatine kinase, Grade 4 | 0
  Creatinine, Grade 1 | 0
  Creatinine, Grade 2 | 0
  Creatinine, Grade 3 | 0
  Creatinine, Grade 4 | 0
  Direct bilirubin, Grade 1 | 0
  Direct bilirubin, Grade 2 | 0
  Direct bilirubin, Grade 3 | 0
  Direct bilirubin, Grade 4 | 0
  GFR from creatinine adjusted using CKD-EPI, Grade 1 | 0
  GFR from creatinine adjusted using CKD-EPI, Grade 2 | 5
  GFR from creatinine adjusted using CKD-EPI, Grade 3 | 1
  GFR from creatinine adjusted using CKD-EPI, Grade 4 | 0
  GFR from creatinine adjusted for BSA, Grade 1 | 0
  GFR from creatinine adjusted for BSA, Grade 2 | 5
  GFR from creatinine adjusted for BSA, Grade 3 | 1
  GFR from creatinine adjusted for BSA, Grade 4 | 0
  Glucose, Grade 1 | 1
  Glucose, Grade 2 | 0
  Glucose, Grade 3 | 0
  Glucose, Grade 4 | 0
  LDL cholesterol calculation, Grade 1 | 0
  LDL cholesterol calculation, Grade 2 | 0
  LDL cholesterol calculation, Grade 3 | 0
  LDL cholesterol calculation, Grade 4 | 0
  Lipase, Grade 1 | 0
  Lipase, Grade 2 | 2
  Lipase, Grade 3 | 0
  Lipase, Grade 4 | 0
  Phosphate, Grade 1 | 0
  Phosphate, Grade 2 | 0
  Phosphate, Grade 3 | 0
  Phosphate, Grade 4 | 0
  Sodium, Grade 1 | 0
  Sodium, Grade 2 | 0
  Sodium, Grade 3 | 0
  Sodium, Grade 4 | 0
  Triglycerides, Grade 1 | 0
  Triglycerides, Grade 2 | 0
  Triglycerides, Grade 3 | 0
  Triglycerides, Grade 4 | 0

20. Secondary Outcome: Number of Participants With Maximum Post-Baseline Hematology Toxicities for CAB LA + RPV LA Q2M Arm up to End of Maintenance Phase
Description: The hematology toxicities were graded as per the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table). Blood samples were collected for the analysis of the hematology parameter: platelets. Severity grades were: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (Potentially life-threatening).
Time Frame: Up to End of Maintenance Phase (up to Month 52)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M
Number analyzed (Participants) | 90
Participants
  Platelets, Grade 1 | 2
  Platelets, Grade 2 | 0
  Platelets, Grade 3 | 0
  Platelets, Grade 4 | 0

21. Secondary Outcome: Number of Participants With Maximum Post-Baseline Hematology Toxicities for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 20
Time Frame: Up to Month 12 [Maintenance Phase]
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Participants
  Platelets, Grade 1 | 0
  Platelets, Grade 2 | 0
  Platelets, Grade 3 | 0
  Platelets, Grade 4 | 0

22. Secondary Outcome: Number of Participants Who Permanently Discontinued Treatment Due to Adverse Events for CAB LA + RPV LA Q2M Arm up to End of Maintenance Phase
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Number of participants with adverse events leading to permanent withdrawal has been presented.
Time Frame: Up to End of Maintenance Phase (up to Month 52)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M
Number analyzed (Participants) | 90
Participants | 1

23. Secondary Outcome: Number of Participants Who Permanently Discontinued Treatment Due to Adverse Events for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 22
Time Frame: Up to Month 12 [Maintenance Phase]
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Participants | 0

24. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatinine Kinase for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemical parameters including ALT, ALP, AST and creatinine kinase. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
International units per liter
  ALT, Month 2: number analyzed (Participants) | 90 | 0
  ALT, Month 2 | -1.1 (16.99) |
  ALT, Month 4: number analyzed (Participants) | 89 | 0
  ALT, Month 4 | -1.0 (26.15) |
  ALT, Month 8: number analyzed (Participants) | 89 | 0
  ALT, Month 8 | 0.0 (29.86) |
  ALT, Month 12: number analyzed (Participants) | 88 | 0
  ALT, Month 12 | 4.0 (44.62) |
  ALT, Month 14: number analyzed (Participants) | 2 | 0
  ALT, Month 14 | -7.5 (61.52) |
  ALT, Month 16: number analyzed (Participants) | 87 | 0
  ALT, Month 16 | -2.5 (24.07) |
  ALT, Month 20: number analyzed (Participants) | 84 | 0
  ALT, Month 20 | -3.4 (18.61) |
  ALT, Month 24: number analyzed (Participants) | 85 | 0
  ALT, Month 24 | -3.0 (17.53) |
  ALT, Month 26: number analyzed (Participants) | 6 | 0
  ALT, Month 26 | -21.7 (49.26) |
  ALT, Month 28: number analyzed (Participants) | 67 | 0
  ALT, Month 28 | 1.0 (31.18) |
  ALT, Month 30: number analyzed (Participants) | 6 | 0
  ALT, Month 30 | 11.2 (49.09) |
  ALT, Month 32: number analyzed (Participants) | 81 | 0
  ALT, Month 32 | -0.9 (18.02) |
  ALT, Month 34: number analyzed (Participants) | 5 | 0
  ALT, Month 34 | -7.0 (30.17) |
  ALT, Month 36: number analyzed (Participants) | 79 | 0
  ALT, Month 36 | 0.2 (18.90) |
  ALT, Month 38: number analyzed (Participants) | 2 | 0
  ALT, Month 38 | 2.5 (4.95) |
  ALT, Month 40: number analyzed (Participants) | 77 | 0
  ALT, Month 40 | -1.7 (19.97) |
  ALT, Month 42: number analyzed (Participants) | 2 | 0
  ALT, Month 42 | -1.5 (6.36) |
  ALT, Month 44: number analyzed (Participants) | 75 | 0
  ALT, Month 44 | -0.5 (14.51) |
  ALT, Month 46: number analyzed (Participants) | 4 | 0
  ALT, Month 46 | 0.5 (3.79) |
  ALT, Month 48: number analyzed (Participants) | 66 | 0
  ALT, Month 48 | -2.6 (11.38) |
  ALT, Month 50: number analyzed (Participants) | 2 | 0
  ALT, Month 50 | -4.5 (7.78) |
  ALT, Month 52: number analyzed (Participants) | 6 | 0
  ALT, Month 52 | -3.5 (13.62) |
  ALT, LTFU Month 1: number analyzed (Participants) | 0 | 5
  ALT, LTFU Month 1 |  | -5.0 (7.07)
  ALT, LTFU Month 3: number analyzed (Participants) | 0 | 4
  ALT, LTFU Month 3 |  | 2.8 (29.93)
  ALT, LTFU Month 6: number analyzed (Participants) | 0 | 6
  ALT, LTFU Month 6 |  | -7.7 (48.87)
  ALT, LTFU Month 9: number analyzed (Participants) | 0 | 6
  ALT, LTFU Month 9 |  | -6.0 (15.17)
  ALT, LTFU Month 12: number analyzed (Participants) | 0 | 5
  ALT, LTFU Month 12 |  | 0.2 (54.36)
  ALP, Month 2: number analyzed (Participants) | 90 | 0
  ALP, Month 2 | 0.2 (8.29) |
  ALP, Month 4: number analyzed (Participants) | 89 | 0
  ALP, Month 4 | 0.2 (14.20) |
  ALP, Month 8: number analyzed (Participants) | 89 | 0
  ALP, Month 8 | 2.0 (11.58) |
  ALP, Month 12: number analyzed (Participants) | 88 | 0
  ALP, Month 12 | 2.1 (12.39) |
  ALP, Month 14: number analyzed (Participants) | 2 | 0
  ALP, Month 14 | -15.5 (33.23) |
  ALP, Month 16: number analyzed (Participants) | 87 | 0
  ALP, Month 16 | 1.7 (10.83) |
  ALP, Month 20: number analyzed (Participants) | 84 | 0
  ALP, Month 20 | 5.5 (11.50) |
  ALP, Month 24: number analyzed (Participants) | 85 | 0
  ALP, Month 24 | 2.3 (12.64) |
  ALP, Month 26: number analyzed (Participants) | 6 | 0
  ALP, Month 26 | -2.2 (23.09) |
  ALP, Month 28: number analyzed (Participants) | 67 | 0
  ALP, Month 28 | 1.0 (12.89) |
  ALP, Month 30: number analyzed (Participants) | 6 | 0
  ALP, Month 30 | 2.3 (19.06) |
  ALP, Month 32: number analyzed (Participants) | 81 | 0
  ALP, Month 32 | 2.4 (11.79) |
  ALP, Month 34: number analyzed (Participants) | 5 | 0
  ALP, Month 34 | 0.4 (10.26) |
  ALP, Month 36: number analyzed (Participants) | 79 | 0
  ALP, Month 36 | 3.3 (9.81) |
  ALP, Month 38: number analyzed (Participants) | 2 | 0
  ALP, Month 38 | -10.0 (14.14) |
  ALP, Month 40: number analyzed (Participants) | 77 | 0
  ALP, Month 40 | 5.7 (14.32) |
  ALP, Month 42: number analyzed (Participants) | 2 | 0
  ALP, Month 42 | 7.0 (2.83) |
  ALP, Month 44: number analyzed (Participants) | 75 | 0
  ALP, Month 44 | 5.3 (16.34) |
  ALP, Month 46: number analyzed (Participants) | 4 | 0
  ALP, Month 46 | 1.8 (7.89) |
  ALP, Month 48: number analyzed (Participants) | 66 | 0
  ALP, Month 48 | 3.3 (12.21) |
  ALP, Month 50: number analyzed (Participants) | 2 | 0
  ALP, Month 50 | 10.5 (2.12) |
  ALP, Month 52: number analyzed (Participants) | 6 | 0
  ALP, Month 52 | -2.5 (7.12) |
  ALP, LTFU Month 1: number analyzed (Participants) | 0 | 5
  ALP, LTFU Month 1 |  | -3.6 (19.24)
  ALP, LTFU Month 3: number analyzed (Participants) | 0 | 4
  ALP, LTFU Month 3 |  | -10.3 (23.91)
  ALP, LTFU Month 6: number analyzed (Participants) | 0 | 6
  ALP, LTFU Month 6 |  | -5.0 (24.71)
  ALP, LTFU Month 9: number analyzed (Participants) | 0 | 6
  ALP, LTFU Month 9 |  | -5.7 (18.28)
  ALP, LTFU Month 12: number analyzed (Participants) | 0 | 5
  ALP, LTFU Month 12 |  | 0.0 (26.31)
  AST, Month 2: number analyzed (Participants) | 90 | 0
  AST, Month 2 | -5.6 (47.9) |
  AST, Month 4: number analyzed (Participants) | 89 | 0
  AST, Month 4 | -5.0 (50.5) |
  AST, Month 8: number analyzed (Participants) | 89 | 0
  AST, Month 8 | -5.3 (49.56) |
  AST, Month 12: number analyzed (Participants) | 88 | 0
  AST, Month 12 | -2.7 (54.93) |
  AST, Month 14: number analyzed (Participants) | 2 | 0
  AST, Month 14 | 0.0 (16.97) |
  AST, Month 16: number analyzed (Participants) | 87 | 0
  AST, Month 16 | -5.1 (51.27) |
  AST, Month 20: number analyzed (Participants) | 84 | 0
  AST, Month 20 | -7.5 (49.83) |
  AST, Month 24: number analyzed (Participants) | 85 | 0
  AST, Month 24 | -7.2 (50.49) |
  AST, Month 26: number analyzed (Participants) | 6 | 0
  AST, Month 26 | -11.5 (15.35) |
  AST, Month 28: number analyzed (Participants) | 67 | 0
  AST, Month 28 | -7.3 (57.53) |
  AST, Month 30: number analyzed (Participants) | 6 | 0
  AST, Month 30 | 3.3 (29.38) |
  AST, Month 32: number analyzed (Participants) | 81 | 0
  AST, Month 32 | -6.7 (51.96) |
  AST, Month 34: number analyzed (Participants) | 5 | 0
  AST, Month 34 | -6.4 (16.56) |
  AST, Month 36: number analyzed (Participants) | 79 | 0
  AST, Month 36 | -5.0 (54.45) |
  AST, Month 38: number analyzed (Participants) | 2 | 0
  AST, Month 38 | -2.0 (7.07) |
  AST, Month 40: number analyzed (Participants) | 77 | 0
  AST, Month 40 | -8.4 (52.46) |
  AST, Month 42: number analyzed (Participants) | 2 | 0
  AST, Month 42 | -0.5 (3.54) |
  AST, Month 44: number analyzed (Participants) | 75 | 0
  AST, Month 44 | -2.0 (9.01) |
  AST, Month 46: number analyzed (Participants) | 4 | 0
  AST, Month 46 | -4.3 (3.59) |
  AST, Month 48: number analyzed (Participants) | 66 | 0
  AST, Month 48 | -3.0 (8.02) |
  AST, Month 50: number analyzed (Participants) | 2 | 0
  AST, Month 50 | -4.5 (3.54) |
  AST, Month 52: number analyzed (Participants) | 6 | 0
  AST, Month 52 | -6.0 (7.90) |
  AST, LTFU Month 1: number analyzed (Participants) | 0 | 5
  AST, LTFU Month 1 |  | 3.6 (18.68)
  AST, LTFU Month 3: number analyzed (Participants) | 0 | 4
  AST, LTFU Month 3 |  | 8.5 (4.51)
  AST, LTFU Month 6: number analyzed (Participants) | 0 | 6
  AST, LTFU Month 6 |  | 1.5 (12.82)
  AST, LTFU Month 9: number analyzed (Participants) | 0 | 6
  AST, LTFU Month 9 |  | 1.5 (6.86)
  AST, LTFU Month 12: number analyzed (Participants) | 0 | 5
  AST, LTFU Month 12 |  | 14.6 (41.38)
  Creatine kinase, Month 2: number analyzed (Participants) | 90 | 0
  Creatine kinase, Month 2 | -255.2 (2327.32) |
  Creatine kinase, Month 4: number analyzed (Participants) | 89 | 0
  Creatine kinase, Month 4 | -204.0 (2483.41) |
  Creatine kinase, Month 8: number analyzed (Participants) | 89 | 0
  Creatine kinase, Month 8 | -237.0 (2362.99) |
  Creatine kinase, Month 12: number analyzed (Participants) | 88 | 0
  Creatine kinase, Month 12 | -252.0 (2429.86) |
  Creatine kinase, Month 14: number analyzed (Participants) | 1 | 0
  Creatine kinase, Month 14 | 120.0 (NA) — Standard Deviation (SD) could not be calculated for a single participant. |
  Creatine kinase, Month 16: number analyzed (Participants) | 87 | 0
  Creatine kinase, Month 16 | -245.1 (2421.43) |
  Creatine kinase, Month 20: number analyzed (Participants) | 84 | 0
  Creatine kinase, Month 20 | -292.8 (2390.38) |
  Creatine kinase, Month 24: number analyzed (Participants) | 85 | 0
  Creatine kinase, Month 24 | -290.0 (2435.94) |
  Creatine kinase, Month 26: number analyzed (Participants) | 6 | 0
  Creatine kinase, Month 26 | -44.0 (115.53) |
  Creatine kinase, Month 28: number analyzed (Participants) | 67 | 0
  Creatine kinase, Month 28 | -393.7 (2738.54) |
  Creatine kinase, Month 30: number analyzed (Participants) | 6 | 0
  Creatine kinase, Month 30 | -33.2 (238.35) |
  Creatine kinase, Month 32: number analyzed (Participants) | 81 | 0
  Creatine kinase, Month 32 | -276.7 (2518.73) |
  Creatine kinase, Month 34: number analyzed (Participants) | 5 | 0
  Creatine kinase, Month 34 | -17.0 (173.27) |
  Creatine kinase, Month 36: number analyzed (Participants) | 79 | 0
  Creatine kinase, Month 36 | -318.6 (2488.91) |
  Creatine kinase, Month 38: number analyzed (Participants) | 2 | 0
  Creatine kinase, Month 38 | -21.0 (32.53) |
  Creatine kinase, Month 40: number analyzed (Participants) | 77 | 0
  Creatine kinase, Month 40 | -341.7 (2552.60) |
  Creatine kinase, Month 42: number analyzed (Participants) | 2 | 0
  Creatine kinase, Month 42 | 30.5 (31.82) |
  Creatine kinase, Month 44: number analyzed (Participants) | 75 | 0
  Creatine kinase, Month 44 | -15.9 (463.41) |
  Creatine kinase, Month 46: number analyzed (Participants) | 4 | 0
  Creatine kinase, Month 46 | 6.0 (50.28) |
  Creatine kinase, Month 48: number analyzed (Participants) | 66 | 0
  Creatine kinase, Month 48 | 1.0 (140.26) |
  Creatine kinase, Month 50: number analyzed (Participants) | 2 | 0
  Creatine kinase, Month 50 | -136.5 (178.90) |
  Creatine kinase, Month 52: number analyzed (Participants) | 6 | 0
  Creatine kinase, Month 52 | -67.7 (84.29) |
  Creatine kinase, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Creatine kinase, LTFU Month 1 |  | -18.0 (21.76)
  Creatine kinase, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Creatine kinase, LTFU Month 3 |  | 81.3 (245.69)
  Creatine kinase, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Creatine kinase, LTFU Month 6 |  | 50.8 (157.89)
  Creatine kinase, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Creatine kinase, LTFU Month 9 |  | -8.8 (88.04)
  Creatine kinase, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Creatine kinase, LTFU Month 12 |  | 844.2 (1731.52)

25. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP, AST and Creatinine Kinase for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 24
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
International units per liter
  ALT, Month 3 | -0.7 (22.37)
  ALT, Month 6 | -4.3 (19.99)
  ALT, Month 9 | 1.7 (8.16)
  ALT, Month 12 | -0.3 (32.32)
  ALP, Month 3 | 1.4 (10.11)
  ALP, Month 6 | 1.6 (8.04)
  ALP, Month 9 | -1.1 (11.74)
  ALP, Month 12 | 10.0 (33.16)
  AST, Month 3 | -0.6 (10.61)
  AST, Month 6 | -3.3 (7.30)
  AST, Month 9 | -1.4 (6.68)
  AST, Month 12 | -0.6 (14.68)
  Creatine kinase, Month 3 | -66.6 (287.66)
  Creatine kinase, Month 6 | -107.9 (112.18)
  Creatine kinase, Month 9 | -90.6 (163.40)
  Creatine kinase, Month 12 | -134.0 (149.59)

26. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Albumin for CAB LA + RPV LA Q2M Arm up to LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemical parameter: albumin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was defined as post-dose visit value minus Baseline value. SD=0.00 is defined as SD resulted below the detectable limit of the assay and approximate to 0.00.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Grams per liter
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | -0.8 (2.31) |
  Month 4: number analyzed (Participants) | 89 | 0
  Month 4 | -0.9 (2.46) |
  Month 8: number analyzed (Participants) | 89 | 0
  Month 8 | -0.8 (2.63) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | -0.9 (2.67) |
  Month 14: number analyzed (Participants) | 1 | 0
  Month 14 | 2.0 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | -0.7 (2.81) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | -0.3 (2.47) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | -0.8 (2.98) |
  Month 26: number analyzed (Participants) | 6 | 0
  Month 26 | 0.8 (2.56) |
  Month 28: number analyzed (Participants) | 67 | 0
  Month 28 | -1.1 (2.68) |
  Month 30: number analyzed (Participants) | 6 | 0
  Month 30 | -0.3 (1.51) |
  Month 32: number analyzed (Participants) | 81 | 0
  Month 32 | -1.2 (2.69) |
  Month 34: number analyzed (Participants) | 5 | 0
  Month 34 | -0.8 (2.68) |
  Month 36: number analyzed (Participants) | 79 | 0
  Month 36 | -1.1 (2.80) |
  Month 38: number analyzed (Participants) | 2 | 0
  Month 38 | -1.0 (1.41) |
  Month 40: number analyzed (Participants) | 77 | 0
  Month 40 | -0.9 (3.00) |
  Month 42: number analyzed (Participants) | 2 | 0
  Month 42 | -3.0 (0.00) |
  Month 44: number analyzed (Participants) | 75 | 0
  Month 44 | -0.9 (2.50) |
  Month 46: number analyzed (Participants) | 4 | 0
  Month 46 | -3.3 (3.50) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | -1.4 (2.56) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -2.5 (2.12) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -1.0 (2.00) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -3.4 (2.88)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | -1.5 (1.29)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -3.0 (3.22)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -2.8 (3.06)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -3.2 (2.05)

27. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Albumin for DTG+ RPV Arm up to Month 12 [Maintenance Phase]
Description: Blood samples were collected for the analysis of clinical chemistry parameter: albumin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Grams per liter
  Month 3 | -1.6 (3.87)
  Month 6 | -1.4 (2.30)
  Month 9 | -1.3 (2.63)
  Month 12 | -2.6 (2.37)

28. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Creatinine for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameters: bilirubin and creatinine. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Micromoles per liter
  Bilirubin, Month 2: number analyzed (Participants) | 90 | 0
  Bilirubin, Month 2 | -1.0 (4.33) |
  Bilirubin, Month 4: number analyzed (Participants) | 89 | 0
  Bilirubin, Month 4 | -1.0 (5.14) |
  Bilirubin, Month 8: number analyzed (Participants) | 89 | 0
  Bilirubin, Month 8 | -1.0 (4.83) |
  Bilirubin, Month 12: number analyzed (Participants) | 88 | 0
  Bilirubin, Month 12 | -0.5 (4.35) |
  Bilirubin, Month 14: number analyzed (Participants) | 2 | 0
  Bilirubin, Month 14 | 2.0 (8.49) |
  Bilirubin, Month 16: number analyzed (Participants) | 87 | 0
  Bilirubin, Month 16 | -1.0 (4.99) |
  Bilirubin, Month 20: number analyzed (Participants) | 84 | 0
  Bilirubin, Month 20 | -1.4 (3.76) |
  Bilirubin, Month 24: number analyzed (Participants) | 85 | 0
  Bilirubin, Month 24 | -0.8 (5.16) |
  Bilirubin, Month 26: number analyzed (Participants) | 6 | 0
  Bilirubin, Month 26 | 0.0 (4.56) |
  Bilirubin, Month 28: number analyzed (Participants) | 67 | 0
  Bilirubin, Month 28 | -0.9 (3.36) |
  Bilirubin, Month 30: number analyzed (Participants) | 6 | 0
  Bilirubin, Month 30 | 2.0 (3.58) |
  Bilirubin, Month 32: number analyzed (Participants) | 81 | 0
  Bilirubin, Month 32 | -1.0 (5.40) |
  Bilirubin, Month 34: number analyzed (Participants) | 5 | 0
  Bilirubin, Month 34 | 0.0 (7.07) |
  Bilirubin, Month 36: number analyzed (Participants) | 79 | 0
  Bilirubin, Month 36 | -0.4 (4.02) |
  Bilirubin, Month 38: number analyzed (Participants) | 2 | 0
  Bilirubin, Month 38 | -2.0 (2.83) |
  Bilirubin, Month 40: number analyzed (Participants) | 77 | 0
  Bilirubin, Month 40 | -1.6 (4.87) |
  Bilirubin, Month 42: number analyzed (Participants) | 2 | 0
  Bilirubin, Month 42 | -1.0 (4.24) |
  Bilirubin, Month 44: number analyzed (Participants) | 75 | 0
  Bilirubin, Month 44 | -0.9 (4.36) |
  Bilirubin, Month 46: number analyzed (Participants) | 4 | 0
  Bilirubin, Month 46 | -3.5 (2.52) |
  Bilirubin, Month 48: number analyzed (Participants) | 66 | 0
  Bilirubin, Month 48 | -1.7 (3.92) |
  Bilirubin, Month 50: number analyzed (Participants) | 2 | 0
  Bilirubin, Month 50 | 1.0 (1.41) |
  Bilirubin, Month 52: number analyzed (Participants) | 6 | 0
  Bilirubin, Month 52 | -1.3 (4.68) |
  Bilirubin, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Bilirubin, LTFU Month 1 |  | -3.2 (5.76)
  Bilirubin, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Bilirubin, LTFU Month 3 |  | 1.5 (7.72)
  Bilirubin, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Bilirubin, LTFU Month 6 |  | 1.3 (9.27)
  Bilirubin, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Bilirubin, LTFU Month 9 |  | 1.0 (9.10)
  Bilirubin, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Bilirubin, LTFU Month 12 |  | -0.8 (6.10)
  Creatinine, Month 2: number analyzed (Participants) | 90 | 0
  Creatinine, Month 2 | -1.84 (7.121) |
  Creatinine, Month 4: number analyzed (Participants) | 89 | 0
  Creatinine, Month 4 | -1.70 (9.393) |
  Creatinine, Month 8: number analyzed (Participants) | 89 | 0
  Creatinine, Month 8 | -0.98 (7.977) |
  Creatinine, Month 10: number analyzed (Participants) | 88 | 0
  Creatinine, Month 10 | -1.14 (9.204) |
  Creatinine, Month 14: number analyzed (Participants) | 1 | 0
  Creatinine, Month 14 | -1.80 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Creatinine, Month 16: number analyzed (Participants) | 87 | 0
  Creatinine, Month 16 | 1.15 (9.508) |
  Creatinine, Month 20: number analyzed (Participants) | 84 | 0
  Creatinine, Month 20 | -0.50 (9.569) |
  Creatinine, Month 24: number analyzed (Participants) | 85 | 0
  Creatinine, Month 24 | 3.57 (10.039) |
  Creatinine, Month 26: number analyzed (Participants) | 6 | 0
  Creatinine, Month 26 | 1.03 (9.423) |
  Creatinine, Month 28: number analyzed (Participants) | 67 | 0
  Creatinine, Month 28 | 4.64 (10.159) |
  Creatinine, Month 30: number analyzed (Participants) | 6 | 0
  Creatinine, Month 30 | 9.87 (8.190) |
  Creatinine, Month 32: number analyzed (Participants) | 81 | 0
  Creatinine, Month 32 | 1.07 (9.648) |
  Creatinine, Month 34: number analyzed (Participants) | 5 | 0
  Creatinine, Month 34 | 1.06 (8.331) |
  Creatinine, Month 36: number analyzed (Participants) | 79 | 0
  Creatinine, Month 36 | 0.76 (9.661) |
  Creatinine, Month 38: number analyzed (Participants) | 3 | 0
  Creatinine, Month 38 | 0.27 (4.007) |
  Creatinine, Month 40: number analyzed (Participants) | 77 | 0
  Creatinine, Month 40 | -2.71 (8.065) |
  Creatinine, Month 42: number analyzed (Participants) | 3 | 0
  Creatinine, Month 42 | 4.73 (7.524) |
  Creatinine, Month 44: number analyzed (Participants) | 76 | 0
  Creatinine, Month 44 | 0.11 (11.223) |
  Creatinine, Month 46: number analyzed (Participants) | 4 | 0
  Creatinine, Month 46 | 8.63 (13.822) |
  Creatinine, Month 48: number analyzed (Participants) | 66 | 0
  Creatinine, Month 48 | 0.01 (9.828) |
  Creatinine, Month 50: number analyzed (Participants) | 2 | 0
  Creatinine, Month 50 | -3.50 (4.950) |
  Creatinine, Month 52: number analyzed (Participants) | 6 | 0
  Creatinine, Month 52 | -2.50 (16.393) |
  Creatinine, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Creatinine, LTFU Month 1 |  | 3.00 (12.761)
  Creatinine, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Creatinine, LTFU Month 3 |  | 13.48 (9.469)
  Creatinine, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Creatinine, LTFU Month 6 |  | 8.42 (12.726)
  Creatinine, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Creatinine, LTFU Month 9 |  | 6.65 (7.731)
  Creatinine, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Creatinine, LTFU Month 12 |  | 9.74 (7.416)

29. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bilirubin, Creatinine for DTG+ RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 28
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Micromoles per liter
  Bilirubin, Month 3 | -1.7 (4.23)
  Bilirubin, Month 6 | -1.4 (3.21)
  Bilirubin, Month 9 | -0.9 (2.54)
  Bilirubin, Month 12 | -1.4 (3.78)
  Creatinine, Month 3 | 11.89 (8.89)
  Creatinine, Month 6 | 8.36 (4.419)
  Creatinine, Month 9 | 16.56 (10.131)
  Creatinine, Month 12 | 7.47 (7.328)

30. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameters: carbon dioxide, chloride, glucose, phosphate, potassium, sodium and urea. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value. SD=0.00(0) is defined as SD resulted below the detectable limit of the assay and approximate to 0.00(0).
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Millimoles per liter
  Carbon dioxide, Month 2: number analyzed (Participants) | 90 | 0
  Carbon dioxide, Month 2 | -0.4 (1.86) |
  Carbon dioxide, Month 4: number analyzed (Participants) | 89 | 0
  Carbon dioxide, Month 4 | -0.1 (2.00) |
  Carbon dioxide, Month 8: number analyzed (Participants) | 89 | 0
  Carbon dioxide, Month 8 | -0.2 (2.22) |
  Carbon dioxide, Month 12: number analyzed (Participants) | 88 | 0
  Carbon dioxide, Month 12 | -0.7 (2.18) |
  Carbon dioxide, Month 14: number analyzed (Participants) | 1 | 0
  Carbon dioxide, Month 14 | 2.0 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Carbon dioxide, Month 16: number analyzed (Participants) | 87 | 0
  Carbon dioxide, Month 16 | 0.3 (2.25) |
  Carbon dioxide, Month 20: number analyzed (Participants) | 84 | 0
  Carbon dioxide, Month 20 | -0.2 (2.17) |
  Carbon dioxide, Month 24: number analyzed (Participants) | 85 | 0
  Carbon dioxide, Month 24 | -0.6 (2.12) |
  Carbon dioxide, Month 26: number analyzed (Participants) | 6 | 0
  Carbon dioxide, Month 26 | 1.7 (3.27) |
  Carbon dioxide, Month 28: number analyzed (Participants) | 67 | 0
  Carbon dioxide, Month 28 | 0.3 (2.61) |
  Carbon dioxide, Month 30: number analyzed (Participants) | 6 | 0
  Carbon dioxide, Month 30 | 1.7 (2.73) |
  Carbon dioxide, Month 32: number analyzed (Participants) | 81 | 0
  Carbon dioxide, Month 32 | 0.4 (2.43) |
  Carbon dioxide, Month 34: number analyzed (Participants) | 5 | 0
  Carbon dioxide, Month 34 | 0.4 (3.13) |
  Carbon dioxide, Month 36: number analyzed (Participants) | 79 | 0
  Carbon dioxide, Month 36 | 0.5 (2.46) |
  Carbon dioxide, Month 38: number analyzed (Participants) | 2 | 0
  Carbon dioxide, Month 38 | 1.0 (1.41) |
  Carbon dioxide, Month 40: number analyzed (Participants) | 77 | 0
  Carbon dioxide, Month 40 | 1.1 (2.63) |
  Carbon dioxide, Month 42: number analyzed (Participants) | 2 | 0
  Carbon dioxide, Month 42 | 0.5 (0.71) |
  Carbon dioxide, Month 44: number analyzed (Participants) | 75 | 0
  Carbon dioxide, Month 44 | 0.7 (2.61) |
  Carbon dioxide, Month 46: number analyzed (Participants) | 4 | 0
  Carbon dioxide, Month 46 | 0.0 (3.74) |
  Carbon dioxide, Month 48: number analyzed (Participants) | 66 | 0
  Carbon dioxide, Month 48 | 0.4 (2.25) |
  Carbon dioxide, Month 50: number analyzed (Participants) | 2 | 0
  Carbon dioxide, Month 50 | 1.0 (2.83) |
  Carbon dioxide, Month 52: number analyzed (Participants) | 6 | 0
  Carbon dioxide, Month 52 | 1.3 (4.32) |
  Carbon dioxide, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Carbon dioxide, LTFU Month 1 |  | 1.0 (3.39)
  Carbon dioxide, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Carbon dioxide, LTFU Month 3 |  | 1.5 (2.52)
  Carbon dioxide, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Carbon dioxide, LTFU Month 6 |  | 0.7 (2.58)
  Carbon dioxide, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Carbon dioxide, LTFU Month 9 |  | 1.0 (2.97)
  Carbon dioxide, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Carbon dioxide, LTFU Month 12 |  | 0.2 (2.28)
  Chloride, Month 2: number analyzed (Participants) | 90 | 0
  Chloride, Month 2 | 1.0 (2.06) |
  Chloride, Month 4: number analyzed (Participants) | 89 | 0
  Chloride, Month 4 | 1.1 (2.20) |
  Chloride, Month 8: number analyzed (Participants) | 89 | 0
  Chloride, Month 8 | 1.2 (2.07) |
  Chloride, Month 12: number analyzed (Participants) | 88 | 0
  Chloride, Month 12 | 1.0 (2.24) |
  Chloride, Month 14: number analyzed (Participants) | 1 | 0
  Chloride, Month 14 | -5.0 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Chloride, Month 16: number analyzed (Participants) | 87 | 0
  Chloride, Month 16 | 0.3 (2.27) |
  Chloride, Month 20: number analyzed (Participants) | 84 | 0
  Chloride, Month 20 | 0.5 (2.52) |
  Chloride, Month 24: number analyzed (Participants) | 85 | 0
  Chloride, Month 24 | 0.3 (2.56) |
  Chloride, Month 26: number analyzed (Participants) | 6 | 0
  Chloride, Month 26 | -2.5 (1.97) |
  Chloride, Month 28: number analyzed (Participants) | 67 | 0
  Chloride, Month 28 | -0.3 (2.42) |
  Chloride, Month 30: number analyzed (Participants) | 6 | 0
  Chloride, Month 30 | -1.7 (2.42) |
  Chloride, Month 32: number analyzed (Participants) | 81 | 0
  Chloride, Month 32 | -0.4 (2.31) |
  Chloride, Month 34: number analyzed (Participants) | 5 | 0
  Chloride, Month 34 | -1.8 (2.28) |
  Chloride, Month 36: number analyzed (Participants) | 79 | 0
  Chloride, Month 36 | -0.5 (2.24) |
  Chloride, Month 38: number analyzed (Participants) | 2 | 0
  Chloride, Month 38 | 1.0 (0.00) |
  Chloride, Month 40: number analyzed (Participants) | 77 | 0
  Chloride, Month 40 | -0.1 (2.40) |
  Chloride, Month 42: number analyzed (Participants) | 2 | 0
  Chloride, Month 42 | -2.0 (4.24) |
  Chloride, Month 44: number analyzed (Participants) | 75 | 0
  Chloride, Month 44 | 0.1 (2.18) |
  Chloride, Month 46: number analyzed (Participants) | 4 | 0
  Chloride, Month 46 | 0.5 (2.65) |
  Chloride, Month 48: number analyzed (Participants) | 66 | 0
  Chloride, Month 48 | -0.3 (2.31) |
  Chloride, Month 50: number analyzed (Participants) | 2 | 0
  Chloride, Month 50 | 0.0 (1.41) |
  Chloride, Month 52: number analyzed (Participants) | 6 | 0
  Chloride, Month 52 | -0.2 (2.32) |
  Chloride, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Chloride, LTFU Month 1 |  | 0.6 (3.91)
  Chloride, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Chloride, LTFU Month 3 |  | -1.8 (3.30)
  Chloride, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Chloride, LTFU Month 6 |  | 0.2 (2.32)
  Chloride, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Chloride, LTFU Month 9 |  | 0.8 (2.14)
  Chloride, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Chloride, LTFU Month 12 |  | -0.2 (2.28)
  Glucose, Month 2: number analyzed (Participants) | 64 | 0
  Glucose, Month 2 | 0.32 (0.568) |
  Glucose, Month 4: number analyzed (Participants) | 62 | 0
  Glucose, Month 4 | 0.42 (0.684) |
  Glucose, Month 8: number analyzed (Participants) | 62 | 0
  Glucose, Month 8 | 0.47 (0.842) |
  Glucose, Month 12: number analyzed (Participants) | 87 | 0
  Glucose, Month 12 | 0.32 (0.662) |
  Glucose, Month 14: number analyzed (Participants) | 1 | 0
  Glucose, Month 14 | -1.60 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Glucose, Month 16: number analyzed (Participants) | 56 | 0
  Glucose, Month 16 | 0.36 (0.754) |
  Glucose, Month 20: number analyzed (Participants) | 56 | 0
  Glucose, Month 20 | 0.33 (0.838) |
  Glucose, Month 24: number analyzed (Participants) | 80 | 0
  Glucose, Month 24 | 0.19 (0.654) |
  Glucose, Month 26: number analyzed (Participants) | 3 | 0
  Glucose, Month 26 | -0.17 (1.457) |
  Glucose, Month 28: number analyzed (Participants) | 48 | 0
  Glucose, Month 28 | 0.30 (0.694) |
  Glucose, Month 30: number analyzed (Participants) | 5 | 0
  Glucose, Month 30 | -0.36 (0.709) |
  Glucose, Month 32: number analyzed (Participants) | 54 | 0
  Glucose, Month 32 | 0.34 (0.792) |
  Glucose, Month 34: number analyzed (Participants) | 2 | 0
  Glucose, Month 34 | 0.95 (2.475) |
  Glucose, Month 36: number analyzed (Participants) | 51 | 0
  Glucose, Month 36 | 0.26 (0.770) |
  Glucose, Month 38: number analyzed (Participants) | 2 | 0
  Glucose, Month 38 | 0.20 (0.566) |
  Glucose, Month 40: number analyzed (Participants) | 49 | 0
  Glucose, Month 40 | 0.25 (0.929) |
  Glucose, Month 42: number analyzed (Participants) | 1 | 0
  Glucose, Month 42 | 0.20 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Glucose, Month 44: number analyzed (Participants) | 48 | 0
  Glucose, Month 44 | 0.54 (1.044) |
  Glucose, Month 46: number analyzed (Participants) | 3 | 0
  Glucose, Month 46 | 0.40 (0.265) |
  Glucose, Month 48: number analyzed (Participants) | 44 | 0
  Glucose, Month 48 | 0.12 (0.593) |
  Glucose, Month 50: number analyzed (Participants) | 2 | 0
  Glucose, Month 50 | 0.40 (0.283) |
  Glucose, Month 52: number analyzed (Participants) | 1 | 0
  Glucose, Month 52 | 2.10 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Glucose, LTFU Month 1: number analyzed (Participants) | 0 | 3
  Glucose, LTFU Month 1 |  | -0.37 (0.058)
  Glucose, LTFU Month 3: number analyzed (Participants) | 0 | 2
  Glucose, LTFU Month 3 |  | -0.45 (0.354)
  Glucose, LTFU Month 6: number analyzed (Participants) | 0 | 4
  Glucose, LTFU Month 6 |  | -0.40 (0.627)
  Glucose, LTFU Month 9: number analyzed (Participants) | 0 | 5
  Glucose, LTFU Month 9 |  | 0.02 (0.259)
  Glucose, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Glucose, LTFU Month 12 |  | -0.12 (0.084)
  Phosphate, Month 2: number analyzed (Participants) | 90 | 0
  Phosphate, Month 2 | -0.00 (0.176) |
  Phosphate, Month 4: number analyzed (Participants) | 89 | 0
  Phosphate, Month 4 | -0.00 (0.191) |
  Phosphate, Month 8: number analyzed (Participants) | 89 | 0
  Phosphate, Month 8 | -0.02 (0.206) |
  Phosphate, Month 12: number analyzed (Participants) | 88 | 0
  Phosphate, Month 12 | -0.02 (0.199) |
  Phosphate, Month 14: number analyzed (Participants) | 1 | 0
  Phosphate, Month 14 | 0.25 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Phosphate, Month 16: number analyzed (Participants) | 87 | 0
  Phosphate, Month 16 | -0.02 (0.199) |
  Phosphate, Month 20: number analyzed (Participants) | 84 | 0
  Phosphate, Month 20 | -0.00 (0.227) |
  Phosphate, Month 24: number analyzed (Participants) | 85 | 0
  Phosphate, Month 24 | -0.01 (0.198) |
  Phosphate, Month 26: number analyzed (Participants) | 6 | 0
  Phosphate, Month 26 | -0.14 (0.206) |
  Phosphate, Month 28: number analyzed (Participants) | 67 | 0
  Phosphate, Month 28 | -0.05 (0.216) |
  Phosphate, Month 30: number analyzed (Participants) | 6 | 0
  Phosphate, Month 30 | 0.05 (0.268) |
  Phosphate, Month 32: number analyzed (Participants) | 81 | 0
  Phosphate, Month 32 | -0.02 (0.186) |
  Phosphate, Month 34: number analyzed (Participants) | 5 | 0
  Phosphate, Month 34 | -0.02 (0.270) |
  Phosphate, Month 36: number analyzed (Participants) | 79 | 0
  Phosphate, Month 36 | -0.01 (0.192) |
  Phosphate, Month 38: number analyzed (Participants) | 2 | 0
  Phosphate, Month 38 | -0.30 (0.212) |
  Phosphate, Month 40: number analyzed (Participants) | 77 | 0
  Phosphate, Month 40 | 0.00 (0.214) |
  Phosphate, Month 42: number analyzed (Participants) | 2 | 0
  Phosphate, Month 42 | 0.10 (0.070) |
  Phosphate, Month 44: number analyzed (Participants) | 75 | 0
  Phosphate, Month 44 | 0.00 (0.201) |
  Phosphate, Month 46: number analyzed (Participants) | 4 | 0
  Phosphate, Month 46 | 0.02 (0.125) |
  Phosphate, Month 48: number analyzed (Participants) | 66 | 0
  Phosphate, Month 48 | 0.01 (0.192) |
  Phosphate, Month 50: number analyzed (Participants) | 2 | 0
  Phosphate, Month 50 | -0.20 (0.141) |
  Phosphate, Month 52: number analyzed (Participants) | 6 | 0
  Phosphate, Month 52 | -0.22 (0.216) |
  Phosphate, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Phosphate, LTFU Month 1 |  | -0.03 (0.222)
  Phosphate, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Phosphate, LTFU Month 3 |  | 0.11 (0.225)
  Phosphate, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Phosphate, LTFU Month 6 |  | -0.02 (0.175)
  Phosphate, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Phosphate, LTFU Month 9 |  | -0.05 (0.165)
  Phosphate, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Phosphate, LTFU Month 12 |  | 0.11 (0.143)
  Potassium, Month 2: number analyzed (Participants) | 90 | 0
  Potassium, Month 2 | 0.06 (0.392) |
  Potassium, Month 4: number analyzed (Participants) | 89 | 0
  Potassium, Month 4 | -0.02 (0.450) |
  Potassium, Month 8: number analyzed (Participants) | 89 | 0
  Potassium, Month 8 | 0.05 (0.408) |
  Potassium, Month 12: number analyzed (Participants) | 88 | 0
  Potassium, Month 12 | 0.06 (0.375) |
  Potassium, Month 14: number analyzed (Participants) | 1 | 0
  Potassium, Month 14 | 0.00 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Potassium, Month 16: number analyzed (Participants) | 87 | 0
  Potassium, Month 16 | 0.00 (0.339) |
  Potassium, Month 20: number analyzed (Participants) | 84 | 0
  Potassium, Month 20 | 0.01 (0.374) |
  Potassium, Month 24: number analyzed (Participants) | 85 | 0
  Potassium, Month 24 | -0.04 (0.384) |
  Potassium, Month 26: number analyzed (Participants) | 6 | 0
  Potassium, Month 26 | 0.10 (0.228) |
  Potassium, Month 28: number analyzed (Participants) | 67 | 0
  Potassium, Month 28 | -0.09 (0.388) |
  Potassium, Month 30: number analyzed (Participants) | 6 | 0
  Potassium, Month 30 | 0.08 (0.293) |
  Potassium, Month 32: number analyzed (Participants) | 81 | 0
  Potassium, Month 32 | 0.00 (0.432) |
  Potassium, Month 34: number analyzed (Participants) | 5 | 0
  Potassium, Month 34 | 0.18 (0.370) |
  Potassium, Month 36: number analyzed (Participants) | 79 | 0
  Potassium, Month 36 | -0.06 (0.411) |
  Potassium, Month 38: number analyzed (Participants) | 2 | 0
  Potassium, Month 38 | 0.35 (0.354) |
  Potassium, Month 40: number analyzed (Participants) | 77 | 0
  Potassium, Month 40 | -0.06 (0.420) |
  Potassium, Month 42: number analyzed (Participants) | 2 | 0
  Potassium, Month 42 | -0.10 (0.424) |
  Potassium, Month 44: number analyzed (Participants) | 75 | 0
  Potassium, Month 44 | -0.04 (0.406) |
  Potassium, Month 46: number analyzed (Participants) | 4 | 0
  Potassium, Month 46 | -0.20 (0.455) |
  Potassium, Month 48: number analyzed (Participants) | 66 | 0
  Potassium, Month 48 | -0.01 (0.374) |
  Potassium, Month 50: number analyzed (Participants) | 2 | 0
  Potassium, Month 50 | 0.00 (0.000) |
  Potassium, Month 52: number analyzed (Participants) | 6 | 0
  Potassium, Month 52 | 0.17 (0.589) |
  Potassium, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Potassium, LTFU Month 1 |  | 0.04 (0.313)
  Potassium, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Potassium, LTFU Month 3 |  | 0.10 (0.606)
  Potassium, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Potassium, LTFU Month 6 |  | 0.13 (0.501)
  Potassium, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Potassium, LTFU Month 9 |  | 0.17 (0.873)
  Potassium, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Potassium, LTFU Month 12 |  | 0.10 (0.212)
  Sodium, Month 2: number analyzed (Participants) | 90 | 0
  Sodium, Month 2 | 0.2 (1.84) |
  Sodium, Month 4: number analyzed (Participants) | 89 | 0
  Sodium, Month 4 | 0.6 (2.10) |
  Sodium, Month 8: number analyzed (Participants) | 89 | 0
  Sodium, Month 8 | 0.6 (1.96) |
  Sodium, Month 12: number analyzed (Participants) | 88 | 0
  Sodium, Month 12 | 0.2 (1.88) |
  Sodium, Month 14: number analyzed (Participants) | 1 | 0
  Sodium, Month 14 | -3.0 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Sodium, Month 16: number analyzed (Participants) | 87 | 0
  Sodium, Month 16 | 0.5 (2.02) |
  Sodium, Month 20: number analyzed (Participants) | 84 | 0
  Sodium, Month 20 | 0.4 (1.96) |
  Sodium, Month 24: number analyzed (Participants) | 85 | 0
  Sodium, Month 24 | 0.5 (1.84) |
  Sodium, Month 26: number analyzed (Participants) | 6 | 0
  Sodium, Month 26 | 0.2 (2.32) |
  Sodium, Month 28: number analyzed (Participants) | 67 | 0
  Sodium, Month 28 | 0.3 (2.12) |
  Sodium, Month 30: number analyzed (Participants) | 6 | 0
  Sodium, Month 30 | -0.8 (2.14) |
  Sodium, Month 32: number analyzed (Participants) | 81 | 0
  Sodium, Month 32 | 0.4 (2.09) |
  Sodium, Month 34: number analyzed (Participants) | 5 | 0
  Sodium, Month 34 | -0.6 (4.72) |
  Sodium, Month 36: number analyzed (Participants) | 79 | 0
  Sodium, Month 36 | -0.1 (2.26) |
  Sodium, Month 38: number analyzed (Participants) | 2 | 0
  Sodium, Month 38 | 1.0 (0.00) |
  Sodium, Month 40: number analyzed (Participants) | 77 | 0
  Sodium, Month 40 | -0.1 (2.11) |
  Sodium, Month 42: number analyzed (Participants) | 2 | 0
  Sodium, Month 42 | -1.0 (1.41) |
  Sodium, Month 44: number analyzed (Participants) | 75 | 0
  Sodium, Month 44 | 0.2 (2.35) |
  Sodium, Month 46: number analyzed (Participants) | 4 | 0
  Sodium, Month 46 | 0.0 (2.94) |
  Sodium, Month 48: number analyzed (Participants) | 66 | 0
  Sodium, Month 48 | 0.1 (1.86) |
  Sodium, Month 50: number analyzed (Participants) | 2 | 0
  Sodium, Month 50 | 1.0 (1.41) |
  Sodium, Month 52: number analyzed (Participants) | 6 | 0
  Sodium, Month 52 | 2.5 (3.15) |
  Sodium, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Sodium, LTFU Month 1 |  | 1.0 (1.22)
  Sodium, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Sodium, LTFU Month 3 |  | -0.5 (1.91)
  Sodium, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Sodium, LTFU Month 6 |  | 0.2 (0.75)
  Sodium, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Sodium, LTFU Month 9 |  | 0.2 (0.75)
  Sodium, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Sodium, LTFU Month 12 |  | -0.4 (0.89)
  Urea, Month 2: number analyzed (Participants) | 90 | 0
  Urea, Month 2 | 0.13 (1.253) |
  Urea, Month 4: number analyzed (Participants) | 89 | 0
  Urea, Month 4 | -0.06 (1.346) |
  Urea, Month 8: number analyzed (Participants) | 89 | 0
  Urea, Month 8 | 0.28 (1.131) |
  Urea, Month 12: number analyzed (Participants) | 88 | 0
  Urea, Month 12 | -0.11 (1.318) |
  Urea, Month 14: number analyzed (Participants) | 1 | 0
  Urea, Month 14 | -0.50 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Urea, Month 16: number analyzed (Participants) | 87 | 0
  Urea, Month 16 | 0.13 (1.444) |
  Urea, Month 20: number analyzed (Participants) | 84 | 0
  Urea, Month 20 | 0.17 (1.332) |
  Urea, Month 24: number analyzed (Participants) | 85 | 0
  Urea, Month 24 | 0.15 (1.474) |
  Urea, Month 26: number analyzed (Participants) | 6 | 0
  Urea, Month 26 | -0.92 (0.736) |
  Urea, Month 28: number analyzed (Participants) | 67 | 0
  Urea, Month 28 | -0.01 (1.628) |
  Urea, Month 30: number analyzed (Participants) | 6 | 0
  Urea, Month 30 | 0.17 (1.941) |
  Urea, Month 32: number analyzed (Participants) | 81 | 0
  Urea, Month 32 | 0.14 (1.419) |
  Urea, Month 34: number analyzed (Participants) | 5 | 0
  Urea, Month 34 | 0.50 (2.000) |
  Urea, Month 36: number analyzed (Participants) | 79 | 0
  Urea, Month 36 | 0.22 (1.393) |
  Urea, Month 38: number analyzed (Participants) | 2 | 0
  Urea, Month 38 | 1.00 (0.707) |
  Urea, Month 40: number analyzed (Participants) | 77 | 0
  Urea, Month 40 | 0.27 (1.390) |
  Urea, Month 42: number analyzed (Participants) | 2 | 0
  Urea, Month 42 | 0.25 (1.061) |
  Urea, Month 44: number analyzed (Participants) | 75 | 0
  Urea, Month 44 | 0.34 (1.475) |
  Urea, Month 46: number analyzed (Participants) | 4 | 0
  Urea, Month 46 | 0.63 (2.056) |
  Urea, Month 48: number analyzed (Participants) | 66 | 0
  Urea, Month 48 | 0.26 (1.266) |
  Urea, Month 50: number analyzed (Participants) | 2 | 0
  Urea, Month 50 | 0.50 (1.414) |
  Urea, Month 52: number analyzed (Participants) | 6 | 0
  Urea, Month 52 | -0.83 (1.211) |
  Urea, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Urea, LTFU Month 1 |  | -0.80 (0.758)
  Urea, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Urea, LTFU Month 3 |  | 0.25 (0.866)
  Urea, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Urea, LTFU Month 6 |  | -1.08 (0.861)
  Urea, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Urea, LTFU Month 9 |  | -0.17 (1.291)
  Urea, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Urea, LTFU Month 12 |  | -0.30 (0.671)

31. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Carbon Dioxide, Chloride, Glucose, Phosphate, Potassium, Sodium and Urea for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: Blood samples were collected for the analysis of clinical chemistry parameters: carbon dioxide, chloride, glucose, phosphate, potassium, sodium and urea. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Millimoles per liter
  Carbon dioxide, Month 3 | -1.0 (1.53)
  Carbon dioxide, Month 6 | -1.7 (1.50)
  Carbon dioxide, Month 9 | -1.9 (2.85)
  Carbon dioxide, Month 12 | -1.9 (2.48)
  Chloride, Month 3 | 1.0 (1.83)
  Chloride, Month 6 | 1.7 (2.14)
  Chloride, Month 9 | 1.0 (0.82)
  Chloride, Month 12 | 1.0 (2.08)
  Glucose, Month 3: number analyzed (Participants) | 5
  Glucose, Month 3 | 0.08 (0.259)
  Glucose, Month 6: number analyzed (Participants) | 5
  Glucose, Month 6 | 0.16 (0.483)
  Glucose, Month 9: number analyzed (Participants) | 4
  Glucose, Month 9 | 0.15 (0.700)
  Glucose, Month 12 | 0.07 (0.55)
  Phosphate, Month 3 | 0.02 (0.131)
  Phosphate, Month 6 | 0.08 (0.177)
  Phosphate, Month 9 | 0.05 (0.178)
  Phosphate, Month 12 | -0.05 (0.101)
  Potassium, Month 3 | -0.26 (0.378)
  Potassium, Month 6 | -0.03 (0.250)
  Potassium, Month 9 | 0.01 (0.135)
  Potassium, Month 12 | -0.06 (0.257)
  Sodium, Month 3 | 0.1 (1.68)
  Sodium, Month 6 | -0.9 (0.90)
  Sodium, Month 9 | -1.0 (2.58)
  Sodium, Month 12 | -1.1 (1.07)
  Urea, Month 3 | 1.43 (0.732)
  Urea, Month 6 | 1.14 (1.144)
  Urea, Month 9 | 1.86 (1.994)
  Urea, Month 12 | 0.71 (0.756)

32. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Cholesterol, High Density Lipoprotein, Cholesterol Direct, Low Density Lipoprotein Cholesterol Calculation, and Cholesterol Direct, Triglycerides for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameters: cholesterol, direct high density lipoprotein cholesterol, LDL cholesterol calculation, direct low density lipoprotein cholesterol and triglycerides. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Millimoles per liter
  Cholesterol, Month 12: number analyzed (Participants) | 88 | 0
  Cholesterol, Month 12 | 0.12 (0.760) |
  Cholesterol, Month 24: number analyzed (Participants) | 85 | 0
  Cholesterol, Month 24 | 0.13 (0.849) |
  Cholesterol, Month 26: number analyzed (Participants) | 6 | 0
  Cholesterol, Month 26 | 0.48 (0.569) |
  Cholesterol, Month 28: number analyzed (Participants) | 35 | 0
  Cholesterol, Month 28 | 0.00 (0.906) |
  Cholesterol, Month 30: number analyzed (Participants) | 2 | 0
  Cholesterol, Month 30 | 0.07 (1.378) |
  Cholesterol, Month 32: number analyzed (Participants) | 2 | 0
  Cholesterol, Month 32 | -0.87 (0.601) |
  Cholesterol, Month 34: number analyzed (Participants) | 2 | 0
  Cholesterol, Month 34 | 0.67 (1.378) |
  Cholesterol, Month 40: number analyzed (Participants) | 3 | 0
  Cholesterol, Month 40 | -0.85 (0.804) |
  Cholesterol, Month 44: number analyzed (Participants) | 2 | 0
  Cholesterol, Month 44 | 0.27 (0.106) |
  Cholesterol, Month 46: number analyzed (Participants) | 1 | 0
  Cholesterol, Month 46 | -0.10 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Cholesterol, Month 48: number analyzed (Participants) | 2 | 0
  Cholesterol, Month 48 | -0.15 (0.070) |
  Cholesterol, LTFU Month 1: number analyzed (Participants) | 0 | 4
  Cholesterol, LTFU Month 1 |  | -0.87 (1.097)
  Cholesterol, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Cholesterol, LTFU Month 12 |  | -0.68 (1.362)
  Direct HDL cholesterol, Month 12: number analyzed (Participants) | 88 | 0
  Direct HDL cholesterol, Month 12 | -0.05 (0.224) |
  Direct HDL cholesterol, Month 24: number analyzed (Participants) | 85 | 0
  Direct HDL cholesterol, Month 24 | -0.02 (0.230) |
  Direct HDL cholesterol, Month 26: number analyzed (Participants) | 6 | 0
  Direct HDL cholesterol, Month 26 | -0.05 (0.154) |
  Direct HDL cholesterol, Month 28: number analyzed (Participants) | 35 | 0
  Direct HDL cholesterol, Month 28 | -0.05 (0.241) |
  Direct HDL cholesterol, Month 30: number analyzed (Participants) | 2 | 0
  Direct HDL cholesterol, Month 30 | 0.25 (0.141) |
  Direct HDL cholesterol, Month 32: number analyzed (Participants) | 2 | 0
  Direct HDL cholesterol, Month 32 | -0.20 (0.353) |
  Direct HDL cholesterol, Month 34: number analyzed (Participants) | 2 | 0
  Direct HDL cholesterol, Month 34 | -0.07 (0.247) |
  Direct HDL cholesterol, Month 40: number analyzed (Participants) | 3 | 0
  Direct HDL cholesterol, Month 40 | 0.08 (0.368) |
  Direct HDL cholesterol, Month 44: number analyzed (Participants) | 2 | 0
  Direct HDL cholesterol, Month 44 | -0.27 (0.247) |
  Direct HDL cholesterol, Month 46: number analyzed (Participants) | 1 | 0
  Direct HDL cholesterol, Month 46 | -0.35 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Direct HDL cholesterol, Month 48: number analyzed (Participants) | 2 | 0
  Direct HDL cholesterol, Month 48 | -0.20 (0.212) |
  Direct HDL cholesterol, LTFU Month 1: number analyzed (Participants) | 0 | 4
  Direct HDL cholesterol, LTFU Month 1 |  | -0.18 (0.213)
  Direct HDL cholesterol, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Direct HDL cholesterol, LTFU Month 12 |  | -0.04 (0.290)
  LDL cholesterol calculation, Month 12: number analyzed (Participants) | 83 | 0
  LDL cholesterol calculation, Month 12 | 0.10 (0.718) |
  LDL cholesterol calculation, Month 24: number analyzed (Participants) | 78 | 0
  LDL cholesterol calculation, Month 24 | 0.14 (0.823) |
  LDL cholesterol calculation, Month 26: number analyzed (Participants) | 5 | 0
  LDL cholesterol calculation, Month 26 | 0.73 (0.613) |
  LDL cholesterol calculation, Month 28: number analyzed (Participants) | 35 | 0
  LDL cholesterol calculation, Month 28 | 0.06 (0.913) |
  LDL cholesterol calculation, Month 30: number analyzed (Participants) | 2 | 0
  LDL cholesterol calculation, Month 30 | 0.31 (2.128) |
  LDL cholesterol calculation, Month 32: number analyzed (Participants) | 2 | 0
  LDL cholesterol calculation, Month 32 | -0.30 (0.502) |
  LDL cholesterol calculation, Month 34: number analyzed (Participants) | 2 | 0
  LDL cholesterol calculation, Month 34 | 0.95 (1.286) |
  LDL cholesterol calculation, Month 40: number analyzed (Participants) | 3 | 0
  LDL cholesterol calculation, Month 40 | -0.91 (0.202) |
  LDL cholesterol calculation, Month 44: number analyzed (Participants) | 2 | 0
  LDL cholesterol calculation, Month 44 | -0.18 (0.530) |
  LDL cholesterol calculation, Month 46: number analyzed (Participants) | 1 | 0
  LDL cholesterol calculation, Month 46 | 0.05 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  LDL cholesterol calculation, Month 48: number analyzed (Participants) | 2 | 0
  LDL cholesterol calculation, Month 48 | -0.03 (0.311) |
  LDL cholesterol calculation, LTFU Month 1: number analyzed (Participants) | 0 | 4
  LDL cholesterol calculation, LTFU Month 1 |  | -0.55 (0.989)
  LDL cholesterol calculation, LTFU Month 12: number analyzed (Participants) | 0 | 5
  LDL cholesterol calculation, LTFU Month 12 |  | -0.34 (1.510)
  Direct LDL cholesterol, Month 12: number analyzed (Participants) | 2 | 0
  Direct LDL cholesterol, Month 12 | 0.21 (0.367) |
  Direct LDL cholesterol, Month 24: number analyzed (Participants) | 1 | 0
  Direct LDL cholesterol, Month 24 | -0.23 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Triglycerides, Month 12: number analyzed (Participants) | 88 | 0
  Triglycerides, Month 12 | 0.28 (1.965) |
  Triglycerides, Month 24: number analyzed (Participants) | 85 | 0
  Triglycerides, Month 24 | 0.20 (1.071) |
  Triglycerides, Month 26: number analyzed (Participants) | 6 | 0
  Triglycerides, Month 26 | -0.20 (0.888) |
  Triglycerides, Month 28: number analyzed (Participants) | 35 | 0
  Triglycerides, Month 28 | -0.02 (0.705) |
  Triglycerides, Month 30: number analyzed (Participants) | 2 | 0
  Triglycerides, Month 30 | -1.06 (1.329) |
  Triglycerides, Month 32: number analyzed (Participants) | 2 | 0
  Triglycerides, Month 32 | -0.80 (0.989) |
  Triglycerides, Month 34: number analyzed (Participants) | 2 | 0
  Triglycerides, Month 34 | -0.43 (0.353) |
  Triglycerides, Month 40: number analyzed (Participants) | 3 | 0
  Triglycerides, Month 40 | -0.04 (1.724) |
  Triglycerides, Month 44: number analyzed (Participants) | 2 | 0
  Triglycerides, Month 44 | 1.61 (0.834) |
  Triglycerides, Month 46: number analyzed (Participants) | 1 | 0
  Triglycerides, Month 46 | 0.44 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Triglycerides, Month 48: number analyzed (Participants) | 2 | 0
  Triglycerides, Month 48 | 0.18 (0.056) |
  Triglycerides, LTFU Month 1: number analyzed (Participants) | 0 | 4
  Triglycerides, LTFU Month 1 |  | -0.29 (0.834)
  Triglycerides, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Triglycerides, LTFU Month 12 |  | -0.64 (1.088)

33. Secondary Outcome: Absolute Values of Clinical Chemistry Parameters: Cholesterol, Direct HDL Cholesterol, LDL Calculation, Direct LDL Cholesterol and Triglycerides for DTG + RPV Arm at Baseline
Description: Blood samples were collected for the analysis of clinical chemistry parameters: cholesterol, HDL cholesterol direct, LDL cholesterol calculation, LDL cholesterol direct and triglycerides.
Time Frame: At Baseline (Day 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Millimoles per liter
  Cholesterol | 4.88 (1.352)
  Direct HDL cholesterol | 1.59 (0.258)
  LDL cholesterol calculation: number analyzed (Participants) | 6
  LDL cholesterol calculation | 2.29 (0.52)
  Direct LDL cholesterol: number analyzed (Participants) | 1
  Direct LDL cholesterol | 4.45 (NA) — Standard deviation could not be calculated for single participant.
  Triglycerides | 1.52 (1.493)

34. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: GFR From Creatinine Adjusted Using CKD-EPI for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: GFR from creatinine adjusted using CKD-EPI. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per minute per 1.73 meter^2
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Milliliter per minute per 1.73 meter^2
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | 1.9 (7.70) |
  Month 4: number analyzed (Participants) | 89 | 0
  Month 4 | 1.7 (10.09) |
  Month 6: number analyzed (Participants) | 5 | 0
  Month 6 | 1.4 (7.86) |
  Month 8: number analyzed (Participants) | 88 | 0
  Month 8 | 0.8 (8.63) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | 0.4 (9.93) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | -1.7 (10.06) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | -0.2 (10.69) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | -5.0 (11.01) |
  Month 26: number analyzed (Participants) | 4 | 0
  Month 26 | 1.8 (5.68) |
  Month 28: number analyzed (Participants) | 48 | 0
  Month 28 | -6.5 (9.44) |
  Month 30: number analyzed (Participants) | 3 | 0
  Month 30 | -12.3 (14.47) |
  Month 32: number analyzed (Participants) | 81 | 0
  Month 32 | -2.1 (9.71) |
  Month 34: number analyzed (Participants) | 4 | 0
  Month 34 | -0.5 (5.07) |
  Month 36: number analyzed (Participants) | 79 | 0
  Month 36 | -2.7 (10.12) |
  Month 38: number analyzed (Participants) | 1 | 0
  Month 38 | -8.0 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Month 40: number analyzed (Participants) | 76 | 0
  Month 40 | 0.8 (8.56) |
  Month 42: number analyzed (Participants) | 3 | 0
  Month 42 | -6.0 (7.94) |
  Month 44: number analyzed (Participants) | 76 | 0
  Month 44 | -1.9 (11.07) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | -8.5 (7.78) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | -2.8 (9.92) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | 2.0 (7.07) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -0.5 (12.85) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -1.2 (9.26)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | -14.3 (10.63)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -10.0 (14.62)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -8.8 (9.87)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -11.0 (7.11)

35. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: GFR From Creatinine Adjusted Using CKD-EPI for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 34
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter per minute per 1.73 meter^2
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Milliliter per minute per 1.73 meter^2
  Month 3 | -11.7 (10.83)
  Month 6 | -7.4 (4.28)
  Month 9 | -16.6 (12.27)
  Month 12 | -7.3 (8.71)

36. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: GFR From Creatinine Adjusted BSA for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: GFR from creatinine adjusted for BSA. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter per second per 1.73 meter^2
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Milliliter per second per 1.73 meter^2
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | 0.03 (0.128) |
  Month 4: number analyzed (Participants) | 89 | 0
  Month 4 | 0.02 (0.168) |
  Month 8: number analyzed (Participants) | 88 | 0
  Month 8 | 0.01 (0.143) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | 0.00 (0.165) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | -0.02 (0.167) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | 0.00 (0.178) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | -0.08 (0.183) |
  Month 26: number analyzed (Participants) | 4 | 0
  Month 26 | 0.02 (0.094) |
  Month 28: number analyzed (Participants) | 48 | 0
  Month 28 | -0.10 (0.157) |
  Month 30: number analyzed (Participants) | 3 | 0
  Month 30 | -0.20 (0.241) |
  Month 32: number analyzed (Participants) | 81 | 0
  Month 32 | -0.03 (0.161) |
  Month 34: number analyzed (Participants) | 4 | 0
  Month 34 | 0.00 (0.084) |
  Month 36: number analyzed (Participants) | 79 | 0
  Month 36 | -0.04 (0.168) |
  Month 38: number analyzed (Participants) | 1 | 0
  Month 38 | -0.13 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Month 40: number analyzed (Participants) | 76 | 0
  Month 40 | 0.01 (0.142) |
  Month 42: number analyzed (Participants) | 3 | 0
  Month 42 | -0.10 (0.132) |
  Month 44: number analyzed (Participants) | 76 | 0
  Month 44 | -0.03 (0.184) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | -0.14 (0.129) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | -0.04 (0.165) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | 0.03 (0.117) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | 0.00 (0.214) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -0.02 (0.154)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | -0.23 (0.177)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -0.16 (0.243)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -0.14 (0.164)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -0.18 (0.118)

37. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: GFR From Creatinine Adjusted BSA for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 36
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter per second per 1.73 meter^2
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Milliliter per second per 1.73 meter^2
  Month 3 | -0.19 (0.180)
  Month 6 | -0.12 (0.071)
  Month 9 | -0.27 (0.204)
  Month 12 | -0.12 (0.145)

38. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Lipase for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: lipase. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Units per liter
  Month 2: number analyzed (Participants) | 90 | 0
  Month 2 | -0.1 (29.11) |
  Month 4: number analyzed (Participants) | 89 | 0
  Month 4 | 3.7 (47.68) |
  Month 6: number analyzed (Participants) | 6 | 0
  Month 6 | 24.5 (64.27) |
  Month 8: number analyzed (Participants) | 89 | 0
  Month 8 | -1.3 (29.43) |
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | -2.9 (36.83) |
  Month 16: number analyzed (Participants) | 87 | 0
  Month 16 | -6.4 (31.83) |
  Month 20: number analyzed (Participants) | 84 | 0
  Month 20 | -4.0 (32.29) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | -2.0 (34.89) |
  Month 26: number analyzed (Participants) | 4 | 0
  Month 26 | 11.0 (4.55) |
  Month 28: number analyzed (Participants) | 48 | 0
  Month 28 | -1.9 (26.19) |
  Month 30: number analyzed (Participants) | 2 | 0
  Month 30 | -1.0 (14.14) |
  Month 32: number analyzed (Participants) | 81 | 0
  Month 32 | 5.5 (56.93) |
  Month 34: number analyzed (Participants) | 4 | 0
  Month 34 | -12.8 (45.17) |
  Month 36: number analyzed (Participants) | 80 | 0
  Month 36 | 4.9 (51.90) |
  Month 38: number analyzed (Participants) | 1 | 0
  Month 38 | 20.0 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Month 40: number analyzed (Participants) | 76 | 0
  Month 40 | 0.7 (41.09) |
  Month 42: number analyzed (Participants) | 3 | 0
  Month 42 | -12.7 (27.39) |
  Month 44: number analyzed (Participants) | 76 | 0
  Month 44 | 5.6 (40.12) |
  Month 46: number analyzed (Participants) | 3 | 0
  Month 46 | -33.3 (118.26) |
  Month 48: number analyzed (Participants) | 66 | 0
  Month 48 | 3.7 (31.55) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -3.0 (28.28) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | 3.2 (12.24) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | 27.4 (48.97)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | 1.5 (10.60)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | 10.8 (30.53)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | 3.7 (9.40)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | 5.2 (6.38)

39. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Lipase for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 38
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Units per liter
  Month 3 | 2.6 (6.90)
  Month 6 | 4.4 (4.35)
  Month 9 | 1.3 (6.85)
  Month 12 | 26.0 (49.76)

40. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Total Cholesterol/ HDL Cholesterol Ratio for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: total cholesterol/ HDL cholesterol ratio. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Total Cholesterol/HDL Cholesterol Ratio
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 88 | 6
Total Cholesterol/HDL Cholesterol Ratio
  Month 12: number analyzed (Participants) | 88 | 0
  Month 12 | 0.20 (1.698) |
  Month 24: number analyzed (Participants) | 85 | 0
  Month 24 | 0.05 (1.279) |
  Month 26: number analyzed (Participants) | 6 | 0
  Month 26 | 0.55 (0.861) |
  Month 28: number analyzed (Participants) | 35 | 0
  Month 28 | 0.11 (1.153) |
  Month 30: number analyzed (Participants) | 2 | 0
  Month 30 | -1.01 (1.630) |
  Month 32: number analyzed (Participants) | 2 | 0
  Month 32 | -0.48 (1.191) |
  Month 34: number analyzed (Participants) | 2 | 0
  Month 34 | 0.43 (0.425) |
  Month 40: number analyzed (Participants) | 3 | 0
  Month 40 | -1.09 (1.390) |
  Month 44: number analyzed (Participants) | 2 | 0
  Month 44 | 1.65 (0.640) |
  Month 46: number analyzed (Participants) | 1 | 0
  Month 46 | 1.37 (NA) — Standard deviation (SD) could not be calculated for a single participant. |
  Month 48: number analyzed (Participants) | 2 | 0
  Month 48 | 0.30 (0.434) |
  LTFU Month 1: number analyzed (Participants) | 0 | 4
  LTFU Month 1 |  | -0.28 (0.916)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -0.51 (1.078)

41. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Total Cholesterol/ HDL Cholesterol Ratio for DTG + RPV Arm at Month 6 [Maintenance Phase]
Description: as for outcome 40
Time Frame: At Month 6 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Total Cholesterol/HDL Cholesterol Ratio
Arm/Group | DTG + RPV
Number analyzed (Participants) | 2
Total Cholesterol/HDL Cholesterol Ratio | 0.55 (0.679)

42. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of hematology parameters: basophils, eosinophils, leukocytes, lymphocytes, monocytes, neutrophils and platelets. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
10^9 cells per liter
  Basophils, Month 2: number analyzed (Participants) | 85 | 0
  Basophils, Month 2 | -0.000 (0.02200) |
  Basophils, Month 4: number analyzed (Participants) | 82 | 0
  Basophils, Month 4 | 0.009 (0.02913) |
  Basophils, Month 8: number analyzed (Participants) | 86 | 0
  Basophils, Month 8 | 0.003 (0.02524) |
  Basophils, Month 12: number analyzed (Participants) | 86 | 0
  Basophils, Month 12 | -0.003 (0.02501) |
  Basophils, Month 16: number analyzed (Participants) | 85 | 0
  Basophils, Month 16 | 0.003 (0.02629) |
  Basophils, Month 20: number analyzed (Participants) | 81 | 0
  Basophils, Month 20 | 0.003 (0.02751) |
  Basophils, Month 22: number analyzed (Participants) | 2 | 0
  Basophils, Month 22 | -0.020 (0.04243) |
  Basophils, Month 24: number analyzed (Participants) | 83 | 0
  Basophils, Month 24 | 0.001 (0.02306) |
  Basophils, Month 26: number analyzed (Participants) | 5 | 0
  Basophils, Month 26 | -0.004 (0.01673) |
  Basophils, Month 28: number analyzed (Participants) | 67 | 0
  Basophils, Month 28 | 0.008 (0.02919) |
  Basophils, Month 30: number analyzed (Participants) | 4 | 0
  Basophils, Month 30 | 0.007 (0.03862) |
  Basophils, Month 32: number analyzed (Participants) | 79 | 0
  Basophils, Month 32 | 0.003 (0.02567) |
  Basophils, Month 34: number analyzed (Participants) | 3 | 0
  Basophils, Month 34 | -0.010 (0.01000) |
  Basophils, Month 36: number analyzed (Participants) | 77 | 0
  Basophils, Month 36 | -0.001 (0.03325) |
  Basophils, Month 38: number analyzed (Participants) | 2 | 0
  Basophils, Month 38 | 0.000 (0.01414) |
  Basophils, Month 40: number analyzed (Participants) | 72 | 0
  Basophils, Month 40 | 0.004 (0.02461) |
  Basophils, Month 42: number analyzed (Participants) | 3 | 0
  Basophils, Month 42 | 0.000 (0.03606) |
  Basophils, Month 44: number analyzed (Participants) | 74 | 0
  Basophils, Month 44 | -0.001 (0.02271) |
  Basophils, Month 46: number analyzed (Participants) | 2 | 0
  Basophils, Month 46 | 0.005 (0.02121) |
  Basophils, Month 48: number analyzed (Participants) | 63 | 0
  Basophils, Month 48 | -0.002 (0.02682) |
  Basophils, Month 50: number analyzed (Participants) | 2 | 0
  Basophils, Month 50 | -0.045 (0.04950) |
  Basophils, Month 52: number analyzed (Participants) | 6 | 0
  Basophils, Month 52 | 0.021 (0.02858) |
  Basophils, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Basophils, LTFU Month 1 |  | 0.004 (0.02702)
  Basophils, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Basophils, LTFU Month 3 |  | 0.000 (0.02944)
  Basophils, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Basophils, LTFU Month 6 |  | -0.001 (0.03764)
  Basophils, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Basophils, LTFU Month 9 |  | 0.000 (0.02000)
  Basophils, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Basophils, LTFU Month 12 |  | 0.010 (0.03240)
  Eosinophils, Month 2: number analyzed (Participants) | 85 | 0
  Eosinophils, Month 2 | 0.017 (0.11886) |
  Eosinophils, Month 4: number analyzed (Participants) | 82 | 0
  Eosinophils, Month 4 | 0.004 (0.12341) |
  Eosinophils, Month 8: number analyzed (Participants) | 86 | 0
  Eosinophils, Month 8 | 0.003 (0.14555) |
  Eosinophils, Month 12: number analyzed (Participants) | 86 | 0
  Eosinophils, Month 12 | -0.000 (0.13671) |
  Eosinophils, Month 16: number analyzed (Participants) | 85 | 0
  Eosinophils, Month 16 | -0.002 (0.12115) |
  Eosinophils, Month 20: number analyzed (Participants) | 81 | 0
  Eosinophils, Month 20 | -0.004 (0.11308) |
  Eosinophils, Month 22: number analyzed (Participants) | 2 | 0
  Eosinophils, Month 22 | 0.005 (0.00707) |
  Eosinophils, Month 24: number analyzed (Participants) | 83 | 0
  Eosinophils, Month 24 | -0.021 (0.10959) |
  Eosinophils, Month 26: number analyzed (Participants) | 5 | 0
  Eosinophils, Month 26 | 0.014 (0.04393) |
  Eosinophils, Month 28: number analyzed (Participants) | 67 | 0
  Eosinophils, Month 28 | -0.021 (0.12165) |
  Eosinophils, Month 30: number analyzed (Participants) | 4 | 0
  Eosinophils, Month 30 | 0.072 (0.09878) |
  Eosinophils, Month 32: number analyzed (Participants) | 79 | 0
  Eosinophils, Month 32 | -0.009 (0.15093) |
  Eosinophils, Month 34: number analyzed (Participants) | 3 | 0
  Eosinophils, Month 34 | 0.083 (0.11846) |
  Eosinophils, Month 36: number analyzed (Participants) | 77 | 0
  Eosinophils, Month 36 | -0.020 (0.13447) |
  Eosinophils, Month 38: number analyzed (Participants) | 2 | 0
  Eosinophils, Month 38 | 0.070 (0.21213) |
  Eosinophils, Month 40: number analyzed (Participants) | 72 | 0
  Eosinophils, Month 40 | -0.014 (0.14536) |
  Eosinophils, Month 42: number analyzed (Participants) | 3 | 0
  Eosinophils, Month 42 | 0.146 (0.04933) |
  Eosinophils, Month 44: number analyzed (Participants) | 74 | 0
  Eosinophils, Month 44 | -0.023 (0.12973) |
  Eosinophils, Month 46: number analyzed (Participants) | 2 | 0
  Eosinophils, Month 46 | 0.065 (0.02121) |
  Eosinophils, Month 48: number analyzed (Participants) | 63 | 0
  Eosinophils, Month 48 | -0.016 (0.13128) |
  Eosinophils, Month 50: number analyzed (Participants) | 2 | 0
  Eosinophils, Month 50 | -0.085 (0.19092) |
  Eosinophils, Month 52: number analyzed (Participants) | 6 | 0
  Eosinophils, Month 52 | -0.020 (0.09675) |
  Eosinophils, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Eosinophils, LTFU Month 1 |  | -0.006 (0.03847)
  Eosinophils, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Eosinophils, LTFU Month 3 |  | -0.042 (0.02062)
  Eosinophils, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Eosinophils, LTFU Month 6 |  | 0.015 (0.05925)
  Eosinophils, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Eosinophils, LTFU Month 9 |  | -0.041 (0.04535)
  Eosinophils, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Eosinophils, LTFU Month 12 |  | 0.036 (0.04930)
  Leukocytes, Month 2: number analyzed (Participants) | 85 | 0
  Leukocytes, Month 2 | -0.054 (1.1875) |
  Leukocytes, Month 4: number analyzed (Participants) | 82 | 0
  Leukocytes, Month 4 | 0.276 (1.4416) |
  Leukocytes, Month 8: number analyzed (Participants) | 86 | 0
  Leukocytes, Month 8 | 0.257 (1.4252) |
  Leukocytes, Month 12: number analyzed (Participants) | 86 | 0
  Leukocytes, Month 12 | -0.153 (1.1961) |
  Leukocytes, Month 16: number analyzed (Participants) | 85 | 0
  Leukocytes, Month 16 | 0.333 (1.4322) |
  Leukocytes, Month 20: number analyzed (Participants) | 81 | 0
  Leukocytes, Month 20 | 0.069 (1.2588) |
  Leukocytes, Month 22: number analyzed (Participants) | 2 | 0
  Leukocytes, Month 22 | -0.050 (0.4950) |
  Leukocytes, Month 24: number analyzed (Participants) | 83 | 0
  Leukocytes, Month 24 | 0.247 (1.3444) |
  Leukocytes, Month 26: number analyzed (Participants) | 5 | 0
  Leukocytes, Month 26 | -0.700 (0.9220) |
  Leukocytes, Month 28: number analyzed (Participants) | 67 | 0
  Leukocytes, Month 28 | 0.369 (1.2534) |
  Leukocytes, Month 30: number analyzed (Participants) | 4 | 0
  Leukocytes, Month 30 | 0.775 (1.1147) |
  Leukocytes, Month 32: number analyzed (Participants) | 79 | 0
  Leukocytes, Month 32 | 0.582 (1.5079) |
  Leukocytes, Month 34: number analyzed (Participants) | 3 | 0
  Leukocytes, Month 34 | -0.033 (0.6351) |
  Leukocytes, Month 36: number analyzed (Participants) | 77 | 0
  Leukocytes, Month 36 | 0.197 (1.3119) |
  Leukocytes, Month 38: number analyzed (Participants) | 2 | 0
  Leukocytes, Month 38 | 0.450 (2.3335) |
  Leukocytes, Month 40: number analyzed (Participants) | 72 | 0
  Leukocytes, Month 40 | 0.111 (1.4863) |
  Leukocytes, Month 42: number analyzed (Participants) | 4 | 0
  Leukocytes, Month 42 | 0.750 (1.6299) |
  Leukocytes, Month 44: number analyzed (Participants) | 74 | 0
  Leukocytes, Month 44 | 0.016 (1.4332) |
  Leukocytes, Month 46: number analyzed (Participants) | 2 | 0
  Leukocytes, Month 46 | 0.700 (0.2828) |
  Leukocytes, Month 48: number analyzed (Participants) | 63 | 0
  Leukocytes, Month 48 | 0.237 (1.3630) |
  Leukocytes, Month 50: number analyzed (Participants) | 2 | 0
  Leukocytes, Month 50 | -2.650 (1.2021) |
  Leukocytes, Month 52: number analyzed (Participants) | 6 | 0
  Leukocytes, Month 52 | 0.950 (0.6804) |
  Leukocytes, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Leukocytes, LTFU Month 1 |  | 0.740 (1.1327)
  Leukocytes, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Leukocytes, LTFU Month 3 |  | 1.100 (1.4720)
  Leukocytes, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Leukocytes, LTFU Month 6 |  | -0.067 (1.0820)
  Leukocytes, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Leukocytes, LTFU Month 9 |  | -0.317 (0.5529)
  Leukocytes, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Leukocytes, LTFU Month 12 |  | -0.240 (0.7369)
  Lymphocytes, Month 2: number analyzed (Participants) | 85 | 0
  Lymphocytes, Month 2 | 0.116 (0.44032) |
  Lymphocytes, Month 4: number analyzed (Participants) | 82 | 0
  Lymphocytes, Month 4 | 0.150 (0.42751) |
  Lymphocytes, Month 8: number analyzed (Participants) | 86 | 0
  Lymphocytes, Month 8 | 0.100 (0.49306) |
  Lymphocytes, Month 12: number analyzed (Participants) | 86 | 0
  Lymphocytes, Month 12 | 0.022 (0.61142) |
  Lymphocytes, Month 16: number analyzed (Participants) | 85 | 0
  Lymphocytes, Month 16 | 0.144 (0.50914) |
  Lymphocytes, Month 20: number analyzed (Participants) | 81 | 0
  Lymphocytes, Month 20 | 0.197 (0.49264) |
  Lymphocytes, Month 22: number analyzed (Participants) | 2 | 0
  Lymphocytes, Month 22 | 0.815 (0.82731) |
  Lymphocytes, Month 24: number analyzed (Participants) | 83 | 0
  Lymphocytes, Month 24 | 0.184 (0.53796) |
  Lymphocytes, Month 26: number analyzed (Participants) | 5 | 0
  Lymphocytes, Month 26 | 0.064 (0.30262) |
  Lymphocytes, Month 28: number analyzed (Participants) | 67 | 0
  Lymphocytes, Month 28 | 0.269 (0.50159) |
  Lymphocytes, Month 30: number analyzed (Participants) | 4 | 0
  Lymphocytes, Month 30 | 0.657 (0.34219) |
  Lymphocytes, Month 32: number analyzed (Participants) | 79 | 0
  Lymphocytes, Month 32 | 0.294 (0.54583) |
  Lymphocytes, Month 34: number analyzed (Participants) | 3 | 0
  Lymphocytes, Month 34 | 0.260 (0.58813) |
  Lymphocytes, Month 36: number analyzed (Participants) | 77 | 0
  Lymphocytes, Month 36 | 0.176 (0.53181) |
  Lymphocytes, Month 38: number analyzed (Participants) | 2 | 0
  Lymphocytes, Month 38 | 0.185 (0.71418) |
  Lymphocytes, Month 40: number analyzed (Participants) | 72 | 0
  Lymphocytes, Month 40 | 0.193 (0.51843) |
  Lymphocytes, Month 42: number analyzed (Participants) | 3 | 0
  Lymphocytes, Month 42 | 0.990 (0.23388) |
  Lymphocytes, Month 44: number analyzed (Participants) | 74 | 0
  Lymphocytes, Month 44 | 0.090 (0.55940) |
  Lymphocytes, Month 46: number analyzed (Participants) | 2 | 0
  Lymphocytes, Month 46 | -0.375 (0.86974) |
  Lymphocytes, Month 48: number analyzed (Participants) | 63 | 0
  Lymphocytes, Month 48 | 0.225 (0.55785) |
  Lymphocytes, Month 50: number analyzed (Participants) | 2 | 0
  Lymphocytes, Month 50 | -0.765 (0.54447) |
  Lymphocytes, Month 52: number analyzed (Participants) | 6 | 0
  Lymphocytes, Month 52 | 0.580 (0.26967) |
  Lymphocytes, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Lymphocytes, LTFU Month 1 |  | 0.316 (0.68995)
  Lymphocytes, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Lymphocytes, LTFU Month 3 |  | 0.215 (0.31268)
  Lymphocytes, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Lymphocytes, LTFU Month 6 |  | 0.018 (0.40276)
  Lymphocytes, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Lymphocytes, LTFU Month 9 |  | -0.013 (0.33339)
  Lymphocytes, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Lymphocytes, LTFU Month 12 |  | 0.182 (0.43906)
  Monocytes, Month 2: number analyzed (Participants) | 85 | 0
  Monocytes, Month 2 | 0.022 (0.11715) |
  Monocytes, Month 4: number analyzed (Participants) | 82 | 0
  Monocytes, Month 4 | 0.048 (0.14689) |
  Monocytes, Month 8: number analyzed (Participants) | 86 | 0
  Monocytes, Month 8 | 0.026 (0.16979) |
  Monocytes, Month 12: number analyzed (Participants) | 86 | 0
  Monocytes, Month 12 | -0.021 (0.15241) |
  Monocytes, Month 16: number analyzed (Participants) | 85 | 0
  Monocytes, Month 16 | 0.060 (0.14219) |
  Monocytes, Month 20: number analyzed (Participants) | 81 | 0
  Monocytes, Month 20 | 0.032 (0.15386) |
  Monocytes, Month 22: number analyzed (Participants) | 2 | 0
  Monocytes, Month 22 | 0.060 (0.11314) |
  Monocytes, Month 24: number analyzed (Participants) | 83 | 0
  Monocytes, Month 24 | 0.039 (0.15115) |
  Monocytes, Month 26: number analyzed (Participants) | 5 | 0
  Monocytes, Month 26 | -0.012 (0.08585) |
  Monocytes, Month 28: number analyzed (Participants) | 67 | 0
  Monocytes, Month 28 | 0.093 (0.15913) |
  Monocytes, Month 30: number analyzed (Participants) | 4 | 0
  Monocytes, Month 30 | 0.105 (0.11328) |
  Monocytes, Month 32: number analyzed (Participants) | 79 | 0
  Monocytes, Month 32 | 0.030 (0.13926) |
  Monocytes, Month 34: number analyzed (Participants) | 3 | 0
  Monocytes, Month 34 | -0.060 (0.06557) |
  Monocytes, Month 36: number analyzed (Participants) | 77 | 0
  Monocytes, Month 36 | 0.016 (0.16850) |
  Monocytes, Month 38: number analyzed (Participants) | 2 | 0
  Monocytes, Month 38 | 0.195 (0.12021) |
  Monocytes, Month 40: number analyzed (Participants) | 72 | 0
  Monocytes, Month 40 | 0.037 (0.17293) |
  Monocytes, Month 42: number analyzed (Participants) | 3 | 0
  Monocytes, Month 42 | 0.230 (0.11358) |
  Monocytes, Month 44: number analyzed (Participants) | 74 | 0
  Monocytes, Month 44 | 0.003 (0.14568) |
  Monocytes, Month 46: number analyzed (Participants) | 2 | 0
  Monocytes, Month 46 | 0.020 (0.08485) |
  Monocytes, Month 48: number analyzed (Participants) | 63 | 0
  Monocytes, Month 48 | 0.026 (0.13077) |
  Monocytes, Month 50: number analyzed (Participants) | 2 | 0
  Monocytes, Month 50 | -0.085 (0.23335) |
  Monocytes, Month 52: number analyzed (Participants) | 6 | 0
  Monocytes, Month 52 | 0.198 (0.13556) |
  Monocytes, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Monocytes, LTFU Month 1 |  | -0.020 (0.06245)
  Monocytes, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Monocytes, LTFU Month 3 |  | -0.007 (0.13451)
  Monocytes, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Monocytes, LTFU Month 6 |  | 0.038 (0.09621)
  Monocytes, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Monocytes, LTFU Month 9 |  | -0.031 (0.09283)
  Monocytes, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Monocytes, LTFU Month 12 |  | 0.008 (0.05541)
  Neutrophils, Month 2: number analyzed (Participants) | 85 | 0
  Neutrophils, Month 2 | -0.197 (0.99349) |
  Neutrophils, Month 4: number analyzed (Participants) | 82 | 0
  Neutrophils, Month 4 | 0.056 (1.19574) |
  Neutrophils, Month 8: number analyzed (Participants) | 86 | 0
  Neutrophils, Month 8 | 0.120 (1.18605) |
  Neutrophils, Month 12: number analyzed (Participants) | 86 | 0
  Neutrophils, Month 12 | -0.134 (1.03311) |
  Neutrophils, Month 16: number analyzed (Participants) | 85 | 0
  Neutrophils, Month 16 | 0.129 (1.23997) |
  Neutrophils, Month 20: number analyzed (Participants) | 81 | 0
  Neutrophils, Month 20 | -0.158 (1.09672) |
  Neutrophils, Month 22: number analyzed (Participants) | 2 | 0
  Neutrophils, Month 22 | -0.890 (1.14551) |
  Neutrophils, Month 24: number analyzed (Participants) | 83 | 0
  Neutrophils, Month 24 | 0.019 (1.06166) |
  Neutrophils, Month 26: number analyzed (Participants) | 5 | 0
  Neutrophils, Month 26 | -0.788 (0.92394) |
  Neutrophils, Month 28: number analyzed (Participants) | 67 | 0
  Neutrophils, Month 28 | 0.025 (1.10870) |
  Neutrophils, Month 30: number analyzed (Participants) | 4 | 0
  Neutrophils, Month 30 | -0.065 (0.70174) |
  Neutrophils, Month 32: number analyzed (Participants) | 79 | 0
  Neutrophils, Month 32 | 0.265 (1.45710) |
  Neutrophils, Month 34: number analyzed (Participants) | 3 | 0
  Neutrophils, Month 34 | -0.310 (0.32187) |
  Neutrophils, Month 36: number analyzed (Participants) | 77 | 0
  Neutrophils, Month 36 | 0.027 (1.15025) |
  Neutrophils, Month 38: number analyzed (Participants) | 2 | 0
  Neutrophils, Month 38 | -0.005 (1.70413) |
  Neutrophils, Month 40: number analyzed (Participants) | 72 | 0
  Neutrophils, Month 40 | -0.100 (1.23231) |
  Neutrophils, Month 42: number analyzed (Participants) | 3 | 0
  Neutrophils, Month 42 | 0.000 (1.35532) |
  Neutrophils, Month 44: number analyzed (Participants) | 74 | 0
  Neutrophils, Month 44 | -0.049 (1.19998) |
  Neutrophils, Month 46: number analyzed (Participants) | 2 | 0
  Neutrophils, Month 46 | 1.015 (1.30815) |
  Neutrophils, Month 48: number analyzed (Participants) | 63 | 0
  Neutrophils, Month 48 | 0.005 (1.16199) |
  Neutrophils, Month 50: number analyzed (Participants) | 2 | 0
  Neutrophils, Month 50 | -1.665 (1.26572) |
  Neutrophils, Month 52: number analyzed (Participants) | 6 | 0
  Neutrophils, Month 52 | 0.151 (0.58952) |
  Neutrophils, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Neutrophils, LTFU Month 1 |  | 0.448 (0.47694)
  Neutrophils, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Neutrophils, LTFU Month 3 |  | 0.932 (1.35866)
  Neutrophils, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Neutrophils, LTFU Month 6 |  | -0.148 (0.90442)
  Neutrophils, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Neutrophils, LTFU Month 9 |  | -0.238 (0.37408)
  Neutrophils, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Neutrophils, LTFU Month 12 |  | -0.462 (0.51611)
  Platelets, Month 2: number analyzed (Participants) | 82 | 0
  Platelets, Month 2 | 3.77 (23.389) |
  Platelets, Month 4: number analyzed (Participants) | 81 | 0
  Platelets, Month 4 | 5.40 (30.889) |
  Platelets, Month 8: number analyzed (Participants) | 84 | 0
  Platelets, Month 8 | 3.74 (24.695) |
  Platelets, Month 12: number analyzed (Participants) | 84 | 0
  Platelets, Month 12 | 1.14 (32.005) |
  Platelets, Month 16: number analyzed (Participants) | 83 | 0
  Platelets, Month 16 | 8.37 (34.613) |
  Platelets, Month 20: number analyzed (Participants) | 78 | 0
  Platelets, Month 20 | 4.19 (33.235) |
  Platelets, Month 22: number analyzed (Participants) | 2 | 0
  Platelets, Month 22 | -10.50 (24.749) |
  Platelets, Month 24: number analyzed (Participants) | 81 | 0
  Platelets, Month 24 | 5.36 (29.747) |
  Platelets, Month 26: number analyzed (Participants) | 4 | 0
  Platelets, Month 26 | 31.00 (34.728) |
  Platelets, Month 28: number analyzed (Participants) | 65 | 0
  Platelets, Month 28 | 7.05 (36.502) |
  Platelets, Month 30: number analyzed (Participants) | 4 | 0
  Platelets, Month 30 | 10.00 (41.873) |
  Platelets, Month 32: number analyzed (Participants) | 77 | 0
  Platelets, Month 32 | 16.29 (43.183) |
  Platelets, Month 34: number analyzed (Participants) | 3 | 0
  Platelets, Month 34 | 24.67 (28.024) |
  Platelets, Month 36: number analyzed (Participants) | 74 | 0
  Platelets, Month 36 | 18.09 (40.388) |
  Platelets, Month 38: number analyzed (Participants) | 2 | 0
  Platelets, Month 38 | 9.50 (38.891) |
  Platelets, Month 40: number analyzed (Participants) | 69 | 0
  Platelets, Month 40 | 12.52 (33.756) |
  Platelets, Month 42: number analyzed (Participants) | 4 | 0
  Platelets, Month 42 | 18.50 (9.434) |
  Platelets, Month 44: number analyzed (Participants) | 72 | 0
  Platelets, Month 44 | 21.07 (40.846) |
  Platelets, Month 46: number analyzed (Participants) | 2 | 0
  Platelets, Month 46 | 28.50 (14.849) |
  Platelets, Month 48: number analyzed (Participants) | 61 | 0
  Platelets, Month 48 | 16.70 (38.627) |
  Platelets, Month 50: number analyzed (Participants) | 2 | 0
  Platelets, Month 50 | -2.50 (7.778) |
  Platelets, Month 52: number analyzed (Participants) | 6 | 0
  Platelets, Month 52 | 22.50 (54.357) |
  Platelets, LTFU Month 1: number analyzed (Participants) | 0 | 5
  Platelets, LTFU Month 1 |  | 10.80 (25.762)
  Platelets, LTFU Month 3: number analyzed (Participants) | 0 | 4
  Platelets, LTFU Month 3 |  | 7.25 (19.973)
  Platelets, LTFU Month 6: number analyzed (Participants) | 0 | 6
  Platelets, LTFU Month 6 |  | -8.00 (24.503)
  Platelets, LTFU Month 9: number analyzed (Participants) | 0 | 6
  Platelets, LTFU Month 9 |  | -13.50 (37.877)
  Platelets, LTFU Month 12: number analyzed (Participants) | 0 | 5
  Platelets, LTFU Month 12 |  | 0.80 (22.709)

43. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 42
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
10^9 cells per liter
  Basophils, Month 3 | -0.008 (0.01464)
  Basophils, Month 6 | -0.010 (0.02309)
  Basophils, Month 9 | -0.005 (0.01512)
  Basophils, Month 12 | -0.010 (0.01732)
  Eosinophils, Month 3 | -0.072 (0.16307)
  Eosinophils, Month 6 | -0.057 (0.11236)
  Eosinophils, Month 9 | -0.051 (0.10040)
  Eosinophils, Month 12 | -0.030 (0.17127)
  Leukocytes, Month 3 | 0.014 (0.7669)
  Leukocytes, Month 6 | -0.386 (0.8355)
  Leukocytes, Month 9 | 0.014 (1.3508)
  Leukocytes, Month 12 | -0.057 (0.9343)
  Lymphocytes, Month 3 | 0.053 (0.43811)
  Lymphocytes, Month 6 | -0.019 (0.35435)
  Lymphocytes, Month 9 | 0.085 (0.59379)
  Lymphocytes, Month 12 | -0.001 (0.39121)
  Monocytes, Month 3 | 0.098 (0.08877)
  Monocytes, Month 6 | 0.020 (0.07211)
  Monocytes, Month 9 | -0.021 (0.06644)
  Monocytes, Month 12 | 0.004 (0.07435)
  Neutrophils, Month 3 | 0.097 (0.47612)
  Neutrophils, Month 6 | -0.295 (0.64143)
  Neutrophils, Month 9 | 0.115 (1.20803)
  Neutrophils, Month 12 | -0.034 (0.80715)
  Platelets, Month 3 | -1.00 (18.841)
  Platelets, Month 6 | -12.57 (35.298)
  Platelets, Month 9 | -21.29 (61.372)
  Platelets, Month 12 | -2.86 (47.544)

44. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Volume for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of hematology parameter: erythrocytes mean corpuscular volume. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Femtoliters
  Month 2: number analyzed (Participants) | 85 | 0
  Month 2 | -1.07 (1.731) |
  Month 4: number analyzed (Participants) | 82 | 0
  Month 4 | -2.04 (2.186) |
  Month 8: number analyzed (Participants) | 86 | 0
  Month 8 | -1.42 (2.527) |
  Month 12: number analyzed (Participants) | 86 | 0
  Month 12 | -1.28 (2.528) |
  Month 16: number analyzed (Participants) | 85 | 0
  Month 16 | -2.91 (2.379) |
  Month 20: number analyzed (Participants) | 81 | 0
  Month 20 | -1.93 (2.544) |
  Month 22: number analyzed (Participants) | 2 | 0
  Month 22 | 2.00 (4.243) |
  Month 24: number analyzed (Participants) | 83 | 0
  Month 24 | -1.35 (2.985) |
  Month 26: number analyzed (Participants) | 5 | 0
  Month 26 | -2.60 (0.894) |
  Month 28: number analyzed (Participants) | 67 | 0
  Month 28 | -3.18 (2.918) |
  Month 30: number analyzed (Participants) | 4 | 0
  Month 30 | -6.75 (2.500) |
  Month 32: number analyzed (Participants) | 79 | 0
  Month 32 | -2.77 (3.355) |
  Month 34: number analyzed (Participants) | 3 | 0
  Month 34 | -3.67 (3.512) |
  Month 36: number analyzed (Participants) | 78 | 0
  Month 36 | -1.78 (2.592) |
  Month 38: number analyzed (Participants) | 2 | 0
  Month 38 | -1.50 (0.707) |
  Month 40: number analyzed (Participants) | 73 | 0
  Month 40 | -3.71 (3.217) |
  Month 42: number analyzed (Participants) | 4 | 0
  Month 42 | -6.75 (2.630) |
  Month 44: number analyzed (Participants) | 74 | 0
  Month 44 | -2.84 (3.167) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | 0.50 (2.121) |
  Month 48: number analyzed (Participants) | 63 | 0
  Month 48 | -2.30 (3.339) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -1.00 (2.828) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -4.00 (3.847) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -3.20 (3.962)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | -4.00 (3.742)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -0.83 (4.167)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -1.33 (4.457)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -1.60 (6.504)

45. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Volume for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 44
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Femtoliters
  Month 3 | -1.00 (1.000)
  Month 6 | 0.14 (1.574)
  Month 9 | 0.29 (1.704)
  Month 12 | -0.14 (1.952)

46. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of hematology parameter: erythrocytes. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value. SD=0.0000 is defined as SD resulted below the detectable limit of the assay and approximate to 0.0000.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
10^12 cells per liter
  Month 2: number analyzed (Participants) | 85 | 0
  Month 2 | -0.064 (0.2773) |
  Month 4: number analyzed (Participants) | 82 | 0
  Month 4 | -0.021 (0.3185) |
  Month 8: number analyzed (Participants) | 86 | 0
  Month 8 | -0.085 (0.3164) |
  Month 12: number analyzed (Participants) | 86 | 0
  Month 12 | -0.063 (0.3279) |
  Month 16: number analyzed (Participants) | 85 | 0
  Month 16 | -0.034 (0.3014) |
  Month 20: number analyzed (Participants) | 81 | 0
  Month 20 | -0.020 (0.2754) |
  Month 22: number analyzed (Participants) | 2 | 0
  Month 22 | -0.450 (0.0707) |
  Month 24: number analyzed (Participants) | 83 | 0
  Month 24 | -0.061 (0.3181) |
  Month 26: number analyzed (Participants) | 5 | 0
  Month 26 | 0.020 (0.1924) |
  Month 28: number analyzed (Participants) | 67 | 0
  Month 28 | -0.113 (0.2949) |
  Month 30: number analyzed (Participants) | 4 | 0
  Month 30 | -0.075 (0.0500) |
  Month 32: number analyzed (Participants) | 79 | 0
  Month 32 | -0.087 (0.3801) |
  Month 34: number analyzed (Participants) | 3 | 0
  Month 34 | -0.233 (0.1155) |
  Month 36: number analyzed (Participants) | 78 | 0
  Month 36 | -0.090 (0.3591) |
  Month 38: number analyzed (Participants) | 2 | 0
  Month 38 | -0.350 (0.3536) |
  Month 40: number analyzed (Participants) | 73 | 0
  Month 40 | -0.056 (0.3528) |
  Month 42: number analyzed (Participants) | 4 | 0
  Month 42 | 0.025 (0.4272) |
  Month 44: number analyzed (Participants) | 74 | 0
  Month 44 | -0.072 (0.4086) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | -0.100 (0.1414) |
  Month 48: number analyzed (Participants) | 63 | 0
  Month 48 | -0.090 (0.3196) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -0.300 (0.0000) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -0.200 (0.5177) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -0.160 (0.2408)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | 0.075 (0.2217)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -0.250 (0.2811)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -0.433 (0.2944)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -0.160 (0.4722)

47. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: Blood samples were collected for the analysis of hematology parameter: erythrocytes. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
10^12 cells per liter
  Month 3 | -0.114 (0.1464)
  Month 6 | -0.171 (0.1113)
  Month 9 | -0.171 (0.1704)
  Month 12 | -0.143 (0.0976)

48. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Proportion of red blood cells in blood
  Month 2: number analyzed (Participants) | 85 | 0
  Month 2 | -0.011 (0.02762) |
  Month 4: number analyzed (Participants) | 82 | 0
  Month 4 | -0.012 (0.02935) |
  Month 8: number analyzed (Participants) | 86 | 0
  Month 8 | -0.015 (0.02809) |
  Month 12: number analyzed (Participants) | 86 | 0
  Month 12 | -0.011 (0.02760) |
  Month 16: number analyzed (Participants) | 85 | 0
  Month 16 | -0.017 (0.02824) |
  Month 20: number analyzed (Participants) | 81 | 0
  Month 20 | -0.011 (0.02731) |
  Month 22: number analyzed (Participants) | 2 | 0
  Month 22 | -0.032 (0.00707) |
  Month 24: number analyzed (Participants) | 83 | 0
  Month 24 | -0.012 (0.02668) |
  Month 26: number analyzed (Participants) | 5 | 0
  Month 26 | -0.010 (0.01723) |
  Month 28: number analyzed (Participants) | 67 | 0
  Month 28 | -0.026 (0.02663) |
  Month 30: number analyzed (Participants) | 4 | 0
  Month 30 | -0.040 (0.00822) |
  Month 32: number analyzed (Participants) | 79 | 0
  Month 32 | -0.022 (0.03499) |
  Month 34: number analyzed (Participants) | 3 | 0
  Month 34 | -0.037 (0.01442) |
  Month 36: number analyzed (Participants) | 78 | 0
  Month 36 | -0.017 (0.03340) |
  Month 38: number analyzed (Participants) | 2 | 0
  Month 38 | -0.034 (0.02192) |
  Month 40: number analyzed (Participants) | 73 | 0
  Month 40 | -0.023 (0.03088) |
  Month 42: number analyzed (Participants) | 4 | 0
  Month 42 | -0.025 (0.03938) |
  Month 44: number analyzed (Participants) | 74 | 0
  Month 44 | -0.021 (0.03702) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | -0.006 (0.00353) |
  Month 48: number analyzed (Participants) | 63 | 0
  Month 48 | -0.019 (0.03114) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -0.033 (0.01697) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -0.041 (0.04229) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -0.028 (0.01864)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | -0.012 (0.02102)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -0.027 (0.03065)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -0.044 (0.02265)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -0.022 (0.03928)

49. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 48
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Proportion of red blood cells in blood
  Month 3 | -0.015 (0.01516)
  Month 6 | -0.013 (0.01287)
  Month 9 | -0.013 (0.01332)
  Month 12 | -0.013 (0.01491)

50. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin for CAB LA + RPV LA Q2M Arm up to End of LTFU Phase
Description: Blood samples were collected for the analysis of hematology parameter: hemoglobin. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: as for outcome 8
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | CAB LA + RPV LA Q2M | LTFU: CAB LA+RPV LA Q2M Group
Number analyzed (Participants) | 90 | 6
Grams per liter
  Month 2: number analyzed (Participants) | 85 | 0
  Month 2 | -2.11 (8.801) |
  Month 4: number analyzed (Participants) | 82 | 0
  Month 4 | -1.57 (9.433) |
  Month 8: number analyzed (Participants) | 86 | 0
  Month 8 | -3.29 (8.542) |
  Month 12: number analyzed (Participants) | 86 | 0
  Month 12 | -3.19 (8.814) |
  Month 16: number analyzed (Participants) | 85 | 0
  Month 16 | -3.44 (8.293) |
  Month 20: number analyzed (Participants) | 81 | 0
  Month 20 | -2.30 (8.054) |
  Month 22: number analyzed (Participants) | 2 | 0
  Month 22 | -13.00 (1.414) |
  Month 24: number analyzed (Participants) | 83 | 0
  Month 24 | -3.35 (8.671) |
  Month 26: number analyzed (Participants) | 5 | 0
  Month 26 | 0.60 (6.804) |
  Month 28: number analyzed (Participants) | 67 | 0
  Month 28 | -4.06 (8.281) |
  Month 30: number analyzed (Participants) | 4 | 0
  Month 30 | -4.00 (4.243) |
  Month 32: number analyzed (Participants) | 79 | 0
  Month 32 | -4.13 (11.183) |
  Month 34: number analyzed (Participants) | 3 | 0
  Month 34 | -8.33 (3.215) |
  Month 36: number analyzed (Participants) | 78 | 0
  Month 36 | -4.86 (10.749) |
  Month 38: number analyzed (Participants) | 2 | 0
  Month 38 | -8.50 (6.364) |
  Month 40: number analyzed (Participants) | 73 | 0
  Month 40 | -4.51 (9.701) |
  Month 42: number analyzed (Participants) | 4 | 0
  Month 42 | -3.50 (11.358) |
  Month 44: number analyzed (Participants) | 74 | 0
  Month 44 | -6.27 (11.766) |
  Month 46: number analyzed (Participants) | 2 | 0
  Month 46 | -6.50 (2.121) |
  Month 48: number analyzed (Participants) | 63 | 0
  Month 48 | -7.41 (9.341) |
  Month 50: number analyzed (Participants) | 2 | 0
  Month 50 | -9.00 (9.899) |
  Month 52: number analyzed (Participants) | 6 | 0
  Month 52 | -6.67 (11.605) |
  LTFU Month 1: number analyzed (Participants) | 0 | 5
  LTFU Month 1 |  | -3.40 (7.956)
  LTFU Month 3: number analyzed (Participants) | 0 | 4
  LTFU Month 3 |  | 1.50 (3.697)
  LTFU Month 6: number analyzed (Participants) | 0 | 6
  LTFU Month 6 |  | -4.67 (9.993)
  LTFU Month 9: number analyzed (Participants) | 0 | 6
  LTFU Month 9 |  | -10.00 (6.000)
  LTFU Month 12: number analyzed (Participants) | 0 | 5
  LTFU Month 12 |  | -1.20 (14.464)

51. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin for DTG + RPV Arm up to Month 12 [Maintenance Phase]
Description: as for outcome 50
Time Frame: At Months 3, 6, 9 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | DTG + RPV
Number analyzed (Participants) | 7
Grams per liter
  Month 3 | -3.57 (6.554)
  Month 6 | -4.29 (2.928)
  Month 9 | -4.86 (3.891)
  Month 12 | -4.57 (5.062)

52. Secondary Outcome: Urine Albumin/Creatinine Ratio and Urine Protein/Creatinine Ratio
Description: Urine samples were collected for the analysis of urine albumin/creatinine ratio and urine protein/creatinine ratio.
Time Frame: At Baseline (Day 1)
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Ratio
  Urine albumin/creatinine ratio: number analyzed (Participants) | 68 | 5
  Urine albumin/creatinine ratio | 0.7 (0.980) | 0.4 (0.122)
  Urine protein/creatinine ratio: number analyzed (Participants) | 73 | 5
  Urine protein/creatinine ratio | 7.6 (4.528) | 9.1 (7.237)

53. Secondary Outcome: Absolute Values of Urine Creatinine
Description: Urine samples were collected for the analysis of urine creatinine.
Time Frame: At Baseline (Day 1)
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Micromoles per liter | 14875.6 (9267.95) | 12112.9 (7186.16)

54. Secondary Outcome: Absolute Values of Urine Phosphate
Description: Urine samples were collected for the analysis of urine phosphate.
Time Frame: At Baseline (Day 1)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Millimoles per liter | 18.2 (15.306) | 14.7 (6.917)

55. Secondary Outcome: Absolute Values of Urine Specific Gravity
Description: Urine samples were collected for the analysis of urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine.
Time Frame: At Baseline (Day 1)
Population: Safety Population. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 89 | 7
Ratio | 1.0 (0.007) | 1.0 (0.007)

56. Secondary Outcome: Absolute Values of Urine Potential of Hydrogen (pH)
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0).
Time Frame: At Baseline (Day 1)
Population: Safety Population. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 89 | 7
pH | 6.1 (0.739) | 6.5 (0.345)

57. Secondary Outcome: Number of Participants With Treatment Emergent Genotypic Resistance
Description: Plasma samples were collected and analyzed for genotypic resistance from participants who met confirmed virologic withdrawal criteria.
Time Frame: Up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase)
Population: Safety Population. Only those participants reporting confirmed virologic failure were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 1 | 0
Participants | 0 |

58. Secondary Outcome: Number of Participants With Treatment Emergent Phenotypic Resistance
Description: Plasma samples were collected and analyzed from participants who met confirmed virologic withdrawal criteria.
Time Frame: Up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase)
Population: Safety Population. Only those participants reporting confirmed virologic failure were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 1 | 0
Participants | 0 |

59. Secondary Outcome: Change From Baseline in HIV Dependent Quality of Life (HIVDQoL - Self-completion Questionnaire Designed to Measure QoL in People Living With HIV)
Description: HIVDQoL includes 2 overview items and 26 domain items. The 2 overview items: Item 1: 3(excellent) to -3(extremely bad); Higher score indicates better quality of life. Item 2: -3(very much better) to 1(worse); Lower score indicates better quality of life. The Weighted Impact Score (WIS) was calculated for the 26 domain items by multiplying impact score(IS) (-3[maximum {max.} negative impact] to +1[max. positive impact] by the corresponding importance score (3 [very important] to 0[not all important]). Average Weighted Impact (AWI) score was calculated by summing individual weighted IS and dividing by the number of domain items. The ranges of WIS and average IS were from -9(max. negative) to +3(max. positive);higher score indicates positive impact. Change from Baseline was defined as post-dose visit value minus Baseline value (latest pre-treatment assessment with a non-missing value). SD=0.00 is defined as SD resulted below the detectable limit of the assay and approximate to 0.00.
Time Frame: At Months 6 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Scores on a scale
  Overview Item 1, Month 6: number analyzed (Participants) | 89 | 7
  Overview Item 1, Month 6 | 0.1 (0.65) | 0.4 (0.53)
  Overview Item 1, Month 12: number analyzed (Participants) | 88 | 7
  Overview Item 1, Month 12 | 0.0 (0.75) | -0.1 (0.38)
  Overview Item 2, Month 6: number analyzed (Participants) | 89 | 7
  Overview Item 2, Month 6 | 0.0 (1.11) | 0.3 (1.25)
  Overview Item 2, Month 12: number analyzed (Participants) | 88 | 7
  Overview Item 2, Month 12 | 0.2 (1.05) | -0.6 (1.13)
  Leisure, Month 6: number analyzed (Participants) | 89 | 7
  Leisure, Month 6 | 0.1 (2.20) | 0.9 (1.46)
  Leisure, Month 12: number analyzed (Participants) | 87 | 7
  Leisure, Month 12 | 0.2 (2.02) | -1.6 (3.74)
  Work, Month 6: number analyzed (Participants) | 86 | 7
  Work, Month 6 | -0.3 (2.07) | -0.9 (4.14)
  Work, Month 12: number analyzed (Participants) | 84 | 7
  Work, Month 12 | -0.1 (2.48) | -0.7 (2.75)
  Holiday, Month 6: number analyzed (Participants) | 84 | 7
  Holiday, Month 6 | -0.5 (2.24) | -0.3 (3.55)
  Holiday, Month 12: number analyzed (Participants) | 84 | 5
  Holiday, Month 12 | -0.1 (2.76) | -2.0 (2.83)
  Getting out and about, Month 6: number analyzed (Participants) | 89 | 7
  Getting out and about, Month 6 | 0.0 (1.83) | -1.1 (3.76)
  Getting out and about, Month 12: number analyzed (Participants) | 88 | 7
  Getting out and about, Month 12 | -0.2 (2.01) | -1.9 (2.48)
  Long journey, Month 6: number analyzed (Participants) | 89 | 7
  Long journey, Month 6 | 0.3 (2.24) | -0.4 (2.70)
  Long journey, Month 12: number analyzed (Participants) | 88 | 7
  Long journey, Month 12 | 0.4 (2.45) | -2.3 (2.93)
  Do Physically, Month 6: number analyzed (Participants) | 89 | 7
  Do Physically, Month 6 | -0.2 (2.09) | -0.7 (2.36)
  Do Physically, Month 12: number analyzed (Participants) | 88 | 7
  Do Physically, Month 12 | -0.3 (2.39) | -1.7 (2.63)
  Family, Month 6: number analyzed (Participants) | 83 | 7
  Family, Month 6 | -0.1 (1.38) | -0.9 (2.27)
  Family, Month 12: number analyzed (Participants) | 82 | 6
  Family, Month 12 | -0.3 (2.30) | -1.5 (2.51)
  Friends, Month 6: number analyzed (Participants) | 89 | 7
  Friends, Month 6 | -0.7 (1.93) | -1.1 (2.85)
  Friends, Month 12: number analyzed (Participants) | 88 | 7
  Friends, Month 12 | -0.3 (2.57) | -2.0 (2.38)
  Go on dates, Month 6: number analyzed (Participants) | 62 | 2
  Go on dates, Month 6 | -0.4 (2.04) | -3.5 (3.54)
  Go on dates, Month 12: number analyzed (Participants) | 60 | 2
  Go on dates, Month 12 | -0.2 (3.11) | -3.5 (3.54)
  Close relationships, Month 6: number analyzed (Participants) | 71 | 6
  Close relationships, Month 6 | 0.4 (3.10) | -0.5 (2.95)
  Close relationships, Month 12: number analyzed (Participants) | 68 | 6
  Close relationships, Month 12 | 0.2 (3.13) | -0.5 (2.95)
  Sex life, Month 6: number analyzed (Participants) | 80 | 6
  Sex life, Month 6 | 0.2 (2.74) | -1.3 (2.80)
  Sex life, Month 12: number analyzed (Participants) | 80 | 5
  Sex life, Month 12 | -0.2 (2.62) | -1.0 (3.00)
  Physical appearance, Month 6: number analyzed (Participants) | 89 | 7
  Physical appearance, Month 6 | -0.3 (1.78) | -1.1 (2.85)
  Physical appearance, Month 12: number analyzed (Participants) | 88 | 7
  Physical appearance, Month 12 | -0.2 (2.28) | -1.4 (2.23)
  Self-confidence, Month 6: number analyzed (Participants) | 88 | 7
  Self-confidence, Month 6 | 0.0 (2.35) | -1.7 (2.43)
  Self-confidence, Month 12: number analyzed (Participants) | 86 | 7
  Self-confidence, Month 12 | 0.2 (2.83) | -2.9 (3.48)
  Motivation, Month 6: number analyzed (Participants) | 89 | 7
  Motivation, Month 6 | -0.3 (2.04) | -0.6 (2.51)
  Motivation, Month 12: number analyzed (Participants) | 86 | 7
  Motivation, Month 12 | -0.3 (2.85) | -2.1 (2.85)
  Stigma, Month 6: number analyzed (Participants) | 40 | 0
  Stigma, Month 6 | -1.1 (2.38) |
  Stigma, Month 12: number analyzed (Participants) | 38 | 1
  Stigma, Month 12 | 0.0 (3.03) | -2.0 (NA) — Standard deviation could not be calculated for single participant.
  Conceal, Month 6: number analyzed (Participants) | 55 | 5
  Conceal, Month 6 | -0.6 (2.91) | -1.6 (3.51)
  Conceal, Month 12: number analyzed (Participants) | 55 | 5
  Conceal, Month 12 | 0.3 (3.04) | -0.4 (4.10)
  Feelings About the Future, Month 6: number analyzed (Participants) | 89 | 7
  Feelings About the Future, Month 6 | 0.0 (2.89) | 1.0 (2.24)
  Feelings About the Future, Month 12: number analyzed (Participants) | 87 | 7
  Feelings About the Future, Month 12 | 0.3 (3.02) | -0.9 (2.85)
  Financial Situation, Month 6: number analyzed (Participants) | 89 | 7
  Financial Situation, Month 6 | -0.1 (2.76) | 1.1 (1.46)
  Financial Situation, Month 12: number analyzed (Participants) | 88 | 7
  Financial Situation, Month 12 | -0.1 (2.59) | -0.6 (4.61)
  Depend on Others, Month 6: number analyzed (Participants) | 37 | 4
  Depend on Others, Month 6 | -0.4 (3.11) | 0.0 (0.00)
  Depend on Others, Month 12: number analyzed (Participants) | 35 | 6
  Depend on Others, Month 12 | -0.2 (2.73) | -1.2 (3.25)
  Others Fuss or Worry, Month 6: number analyzed (Participants) | 42 | 5
  Others Fuss or Worry, Month 6 | 0.0 (3.00) | -1.6 (3.36)
  Others Fuss or Worry, Month 12: number analyzed (Participants) | 35 | 6
  Others Fuss or Worry, Month 12 | 0.1 (3.21) | -0.3 (3.50)
  Freedom to Eat, Month 6: number analyzed (Participants) | 89 | 7
  Freedom to Eat, Month 6 | 0.0 (1.98) | -1.3 (3.40)
  Freedom to Eat, Month 12: number analyzed (Participants) | 88 | 7
  Freedom to Eat, Month 12 | 0.1 (2.62) | -1.1 (2.48)
  Freedom to Drink, Month 6: number analyzed (Participants) | 88 | 7
  Freedom to Drink, Month 6 | -0.2 (1.81) | -0.7 (4.42)
  Freedom to Drink, Month 12: number analyzed (Participants) | 87 | 7
  Freedom to Drink, Month 12 | -0.1 (2.47) | -1.7 (3.40)
  Spiritual/Religious Life, Month 6: number analyzed (Participants) | 46 | 6
  Spiritual/Religious Life, Month 6 | -0.1 (2.46) | -0.5 (1.22)
  Spiritual/Religious Life, Month 12: number analyzed (Participants) | 45 | 6
  Spiritual/Religious Life, Month 12 | -0.1 (1.14) | -1.0 (2.45)
  Feelings About the Past, Month 6: number analyzed (Participants) | 88 | 7
  Feelings About the Past, Month 6 | -0.3 (2.69) | 0.7 (2.21)
  Feelings About the Past, Month 12: number analyzed (Participants) | 87 | 7
  Feelings About the Past, Month 12 | 0.0 (2.74) | -1.3 (2.21)
  Having Children or More Children, Month 6: number analyzed (Participants) | 30 | 4
  Having Children or More Children, Month 6 | 0.3 (1.86) | 1.3 (4.27)
  Having Children or More Children, Month 12: number analyzed (Participants) | 35 | 4
  Having Children or More Children, Month 12 | -0.3 (2.82) | -1.5 (3.00)
  Sleep, Month 6: number analyzed (Participants) | 87 | 7
  Sleep, Month 6 | -0.2 (2.32) | 0.7 (1.25)
  Sleep, Month 12: number analyzed (Participants) | 87 | 7
  Sleep, Month 12 | 0.0 (2.56) | -0.4 (2.70)
  Average Weighted Impact, Month 6: number analyzed (Participants) | 89 | 7
  Average Weighted Impact, Month 6 | -0.17 (1.084) | -0.43 (1.792)
  Average Weighted Impact, Month 12: number analyzed (Participants) | 88 | 7
  Average Weighted Impact, Month 12 | -0.07 (1.690) | -1.27 (1.695)

60. Secondary Outcome: Change From Baseline in Total Treatment Satisfaction Score of HIV Treatment Satisfaction Status Questionnaire (HIVTSQs)
Description: HIVTSQs total treatment satisfaction score is computed with 1-11 items. Items 1-11 are summed to produce score with possible range of 0 to 66. Higher the score, greater improvement in satisfaction with treatment as compared to the past few weeks; lower score, greater the deterioration in satisfaction with treatment. A score of 0 represents no change. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. Change from baseline was defined as post-dose visit value minus baseline value.
Time Frame: At Months 6 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Scores on a scale
  Month 6: number analyzed (Participants) | 89 | 7
  Month 6 | -0.19 (6.419) | 0.71 (3.773)
  Month 12: number analyzed (Participants) | 88 | 7
  Month 12 | -0.42 (6.659) | 0.14 (6.256)

61. Secondary Outcome: Change From Baseline in Individual Item Score of HIVTSQs
Description: HIVTSQs is a 12 item questionnaire. The individual item scores are rated as 6 (very satisfied, convenient, flexible, etc.) to 0 (very dissatisfied, inconvenient, inflexible, etc.). Higher scores represent greater treatment satisfaction as compared to the past few weeks. Change from Baseline is defined as post-dose value minus Baseline value. Baseline value is defined as latest pre-treatment assessment with a non-missing value, including those from unscheduled visits. SD=0.00 is defined as SD resulted below the detectable limit of the assay and approximate to 0.00.
Time Frame: At Months 6 and 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 90 | 7
Scores on a scale
  Item 1, Month 6: number analyzed (Participants) | 89 | 7
  Item 1, Month 6 | -0.1 (0.82) | 0.0 (0.00)
  Item 1, Month 12: number analyzed (Participants) | 88 | 7
  Item 1, Month 12 | -0.1 (0.75) | -0.1 (0.38)
  Item 2, Month 6: number analyzed (Participants) | 89 | 7
  Item 2, Month 6 | -0.1 (0.46) | -0.3 (0.49)
  Item 2, Month 12: number analyzed (Participants) | 88 | 7
  Item 2, Month 12 | 0.0 (0.34) | -0.1 (0.38)
  Item 3, Month 6: number analyzed (Participants) | 89 | 7
  Item 3, Month 6 | -0.5 (1.41) | 0.1 (0.38)
  Item 3, Month 12: number analyzed (Participants) | 88 | 7
  Item 3, Month 12 | -0.5 (1.21) | -0.1 (0.38)
  Item 4, Month 6: number analyzed (Participants) | 89 | 7
  Item 4, Month 6 | 0.0 (0.95) | 0.0 (0.00)
  Item 4, Month 12: number analyzed (Participants) | 88 | 7
  Item 4, Month 12 | 0.1 (0.93) | 0.1 (0.69)
  Item 5, Month 6: number analyzed (Participants) | 89 | 7
  Item 5, Month 6 | 0.1 (1.00) | 0.3 (0.49)
  Item 5, Month 12: number analyzed (Participants) | 87 | 7
  Item 5, Month 12 | 0.1 (1.14) | 0.1 (0.38)
  Item 6, Month 6: number analyzed (Participants) | 88 | 7
  Item 6, Month 6 | 0.1 (1.13) | 0.4 (1.62)
  Item 6, Month 12: number analyzed (Participants) | 88 | 7
  Item 6, Month 12 | 0.0 (1.31) | 0.3 (1.80)
  Item 7, Month 6: number analyzed (Participants) | 89 | 7
  Item 7, Month 6 | 0.1 (0.74) | 0.0 (0.58)
  Item 7, Month 12: number analyzed (Participants) | 88 | 7
  Item 7, Month 12 | 0.0 (1.06) | 0.1 (0.69)
  Item 8, Month 6: number analyzed (Participants) | 89 | 7
  Item 8, Month 6 | 0.2 (0.93) | 0.0 (0.58)
  Item 8, Month 12: number analyzed (Participants) | 88 | 7
  Item 8, Month 12 | 0.1 (0.95) | 0.0 (0.58)
  Item 9, Month 6: number analyzed (Participants) | 89 | 7
  Item 9, Month 6 | -0.1 (0.61) | 0.0 (0.00)
  Item 9, Month 12: number analyzed (Participants) | 88 | 7
  Item 9, Month 12 | -0.2 (0.80) | -0.1 (0.38)
  Item 10, Month 6: number analyzed (Participants) | 89 | 7
  Item 10, Month 6 | 0.1 (0.91) | 0.3 (0.76)
  Item 10, Month 12: number analyzed (Participants) | 88 | 7
  Item 10, Month 12 | 0.1 (1.03) | 0.1 (0.90)
  Item 11, Month 6: number analyzed (Participants) | 89 | 7
  Item 11, Month 6 | 0.0 (1.09) | -0.1 (0.38)
  Item 11, Month 12: number analyzed (Participants) | 88 | 7
  Item 11, Month 12 | 0.1 (0.79) | -0.1 (0.90)
  Item 12, Month 6: number analyzed (Participants) | 89 | 7
  Item 12, Month 6 | -1.3 (1.59) | -0.6 (1.13)
  Item 12, Month 12: number analyzed (Participants) | 88 | 7
  Item 12, Month 12 | -1.1 (1.58) | -0.1 (0.38)

62. Secondary Outcome: Change in Treatment Satisfaction Over Time Using the HIV Treatment Satisfaction Change Questionnaire (HIVTSQc)
Description: HIVTSQc (change version) total treatment satisfaction score is computed with 1-11 items. Items 1-11 are summed to produce score with possible range:-33 to 33. Higher scores represent greater improvement in treatment satisfaction compared to satisfaction with treatment received during the induction phase; lower scores represented deterioration in satisfaction with treatment. A score of 0 represents no change. A maximum of 5 items can be missing, the missing scores were imputed with the mean of the completed item scores. If 6 or more items are missing, then the overall treatment satisfaction scale score was not computed and remained missing.
Time Frame: At Month 12 (compared with Baseline [Day 1]) [Maintenance Phase]
Population: ITT-E Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV
Number analyzed (Participants) | 88 | 7
Scores on a scale | 28.0 (6.78) | 27.7 (6.97)

63. Other Pre Specified Outcome: Plasma Trough Concentration (Ctrough) for CAB LA
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of CAB LA. This was a conditional secondary endpoint for which results are not available because the trough concentrations for this product are well characterized and therefore, secondary population pharmacokinetic (Pop PK) analyses were not conducted.
Time Frame: Pre-dose (Day 1) and Month 12 [Maintenance Phase]
Population: Pharmacokinetic Population
Groups:
- CAB LA: Participants in this arm received their first dose CAB LA (600 mg) injection within 2 hours of the final oral dose of LATTE given on the same day. The second loading injections were administered 1 month after initial loading dose, with subsequent injection (CAB LA 600 mg) occurring Q2M thereafter.
Arm/Group | CAB LA
Number analyzed (Participants) | 0

64. Other Pre Specified Outcome: Ctrough for RPV LA
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of RPV LA. This was a conditional secondary endpoint for which results are not available because the trough concentrations for this product are well characterized and therefore, secondary Pop PK analyses were not conducted.
Time Frame: Pre-dose (Day 1) and Month 12 [Maintenance Phase]
Population: Pharmacokinetic Population
Groups:
- RPV LA: Participants in this arm received their first dose RPV LA (900 mg) injection within 2 hours of the final oral dose of LATTE given on the same day. The second loading injections were administered 1 month after initial loading dose, with subsequent injection (RPV LA 900 mg) occurring Q2M thereafter.
Arm/Group | RPV LA
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Non-Serious adverse events (Other Adverse events (AEs)) and Serious adverse events (SAE) were collected from Day 1 and up to End of LTFU Phase (approximately up to 12 months after exiting the Maintenance Phase, up to a maximum of 52 months).
Description: As specified in protocol, Non-SAEs (Other AEs) and SAEs were only collected on participants who received at least one dose of study treatment on or after Day 1 visit.
Arm/Group | CAB LA + RPV LA Q2M | DTG + RPV | LTFU: CAB LA+RPV LA Q2M Group
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 10/90 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 86/90 | 3/7 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA + RPV LA Q2M (N=90) | DTG + RPV (N=7) | LTFU: CAB LA+RPV LA Q2M Group (N=6)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAB LA + RPV LA Q2M (N=90) | DTG + RPV (N=7) | LTFU: CAB LA+RPV LA Q2M Group (N=6)
Injection site pain (General disorders) | 67 (699) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 13 (31) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 14 (36) | 0 (0) | 0 (0)
Fatigue (General disorders) | 11 (34) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 10 (18) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 7 (14) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 14 (14) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (24) | 0 (0) | 0 (0)
Syphilis (Infections and infestations) | 13 (19) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (20) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 8 (8) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (15) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 7 (9) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 6 (12) | 0 (0) | 0 (0)
Pain (General disorders) | 6 (13) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 5 (7) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 30 (33) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 6 (7) | 0 (0) | 0 (0)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 7 (7) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 10 (11) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03639311/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT03639311/SAP_001.pdf